

# Statistical Analysis Plan

jCyte, Inc. Protocol JC-01

A Prospective, Multicenter, Open-Label, Single-Arm Study of the Safety and Tolerability of a Single, Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects with Retinitis Pigmentosa (RP)

Protocol Version: Amendment 6 (July 07, 2016)

**Sponsor:** jCyte, Inc

2549 East bluff Drive, Suite 196 Newport Beach, CA 92660

Prepared by: Suma Bojadlaa

SynteractHCR, Inc. 5759 Fleet Street Carlsbad, CA 92008

| Version | Date |
|------------|------------|
| Final V1.0 | 19 Jul2017 |
| Final V2.0 | 08Nov2017 |

# Approval

Upon review of this document, including table, listing, and figure shells, the undersigned approves the Statistical Analysis Plan. The analysis methods and data presentation are acceptable.

| Signature | | ate |
|---|---|---|
| Hospiethan, Morra (Bown, Ambriega) Hospiethan, Morra (Bown, Ambriega) Brown of 2017 (1991) at 100 1000 COSSSS 1 | | |
| Suma Bojadlaa, MS | <u>~</u> | <u> </u> |
| Biostatistician II | | × |
| 5 Synteract | - 000/750 | |
| Amarya, Ramesh Dieckur, Biotachistica Tomore the document 08 New 2017 13:52:59-48:90 | cosign | |
| Ramesh Amatya, PhD | _ | <del></del> |
| Director, Biostatistics | | |
| 5 Synteract | | |
| Bound Nills | | 11/8/17 |
| Mills Bonnie | - | 7 7 ( |
| Consultant to jcyte | | |
| jCyte, Inc. | | |

# TABLE OF CONTENTS

| LIS | T OF | ABBREVIATIONS | 5 |
|-----|-------|------------------------------------------|------|
| DE | FINIT | TONS | 8 |
| 1. | INTE | RODUCTION | 9 |
| 2. | STU | DY OBJECTIVES | 9 |
| | 2.1 P | RIMARY OBJECTIVE | 9 |
| | | ECONDARY OBJECTIVE | |
| 3. | STU | DY DESIGN AND PLAN | 9 |
| 4. | DET | ERMINATION OF SAMPLE SIZE | . 11 |
| 5. | | ERAL ANALYSIS CONSIDERATIONS | |
| 6. | | LYSIS POPULATIONS | |
| 7. | | DY POPULATION | |
| | 7.1 | SUBJECT DISPOSITION | |
| | 7.2 | PROTOCOL DEVIATIONS | |
| | 7.3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | . 13 |
| | 7.4 | PRIOR AND CONCOMITANT MEDICATIONS | . 14 |
| 8. | EFFI | ICACY ANALYSES | . 14 |
| | 8.1 | EFFICACY VARIABLES | . 14 |
| | 8.2 | BASELINE VALUES | |
| | 8.3 | HANDLING OF DROPOUTS OR MISSING DATA | |
| | 8.4 | INTERIM ANALYSIS AND DATA MONITORING | |
| | 8.5 | EXAMINATION OF SUBGROUPS | |
| | 8.6 | MULTIPLE COMPARISON/MULTIPLICITY | |
| | 8.7 | MULTICENTER STUDIES | . 16 |
| 9. | MET | THODS OF EFFICACY ANALYSIS | . 16 |
| | 9.1 | BEST CORRECTED VISUAL ACUITY (BCVA) | . 16 |
| | 9.2 | ELECTRORETINOGRAM (ERG) | . 17 |
| | 9.3 | VISUAL FIELD EXAMINATION | |
| 10. | SAFI | ETY ANALYSES | . 17 |
| | 10.1 | STUDY DRUG ADMINISTRATION | . 18 |
| | 10.2 | ADVERSE EVENTS | . 18 |
| | | CLINICAL LABORATORY EVALUATION | |
| | 10.4 | VITAL SIGNS | |
| | 10.5 | PHYSICAL EXAMINATION | |
| | 10.6 | ELECTROCARDIOGRAM | |
| | | OPHTHALMIC AES | |
| | | 1 SLIT LAMP AND FUNDUS PHOTOGRAPHY | |
| | 10.7. | 2 Intraocular Pressure (IOP) | . 20 |

| | 10.7.3 B-SCAN | 20 |
|-----|-----------------------------------------------------------------|----|
| | 10.7.4 DILATED FUNDOSCOPIC EXAMINATION | 21 |
| | 10.7.5 Post Injection Clinical Vitreous Exam | 21 |
| | 10.7.6 OPTICAL COHERENCE TOMOGRAPHY (OCT) | |
| | 10.7.7FLUORESCEIN ANGIOGRAPHY | |
| | 10.7.8 AUTOFLUORESCENCE | 21 |
| 11. | REFERENCES | 21 |
| | APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS | 23 |
| | APPENDIX B: LIST OF TABLES, FIGURES, AND LISTINGS | 26 |
| | APPENDIX C: TABLE LAYOUTS | |
| | ADDENDIN D. LICTING LANGUES | 70 |

#### LIST OF ABBREVIATIONS

AE Adverse Event

ATC Anatomical Therapeutic Chemical

BCVA Best Corrected Visual Acuity

BP Blood Pressure
bpm Beats per Minute
cm Centimeter(s)
CRF Case Report Form
CS Clinically Significant
CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

DDT Dictionary Derived Term

ECG Electrocardiogram

E-ETDRS Electronic Early Treatment for Diabetic Retinopathy Study

ERG Electroretinogram EZ Ellipsoid Zone

hRPC Human Retinal Progenitor Cells

ICH International Conference on Harmonization

in Inch(es)

ITT Intent-to-Treat kg kilogram(s) msec Millisecond

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram(s)

mmHg Millimeter of Mercury NCS Not Clinically Significant

OCT Optical Coherence Tomography
OD Oculus Dextrus (right eye)
OS Oculus Sinister (left eye)

PT Preferred Term

QTc Corrected QT Interval

QTcB Corrected QT Interval According to Bazett's formula
QTcF Corrected QT Interval According to Fridericia's formula

# LIST OF ABBREVIATIONS (continued)

| RP | Retinitis Pigmentosa |
|-----|---------------------------|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |

TEAE Treatment-Emergent Adverse Event

TLs Tables and Listings

VFQ-25 Visual Function Questionnaire WHO World Health Organization

### **DEFINITIONS**

Adverse Event An adverse event (AE) is any reaction, side effect, or

other untoward event, regardless of relationship to study

drug, which occurs anytime during the study.

All subjects who enroll in the study and who provide any Intent-to-Treat Population

post-screening data

Safety Population

All subjects who received any amount of study drug Serious AE An AE occurring at any dose that: results in death; is a

> life-threatening experience; requires inpatient hospitalization or prolongation of an existing hospitalization; results in a persistent or significant disability/incapacity; or is a congenital anomaly/birth defect in the offspring of a subject who received study

drug.

AEs with an onset time after the initial dose of study Treatment-emergent AE

drug.

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of jCyte Protocol JC-01 [A Prospective, Multicenter, Open-Label, Single -Arm Study of the Safety and Tolerability of a Single, Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects with Retinitis Pigmentosa (RP)]. The purpose of this plan is to provide specific guidelines from which the statistical analyses will proceed. Any deviations from this plan will be documented in the clinical study report (CSR).

#### 2. STUDY OBJECTIVES

# 2.1 Primary Objective

The primary objective is to evaluate the safety and tolerability of jCell injection in adult subjects with non-syndromic RP.

# 2.2 Secondary Objective

The secondary objectives of the study are to monitor ocular function over a 12 month period following a single injection of hRPC (jCell) to evaluate the potential therapeutic response in subjects with RP.

### 3. STUDY DESIGN AND PLAN

This is a prospective, multicenter, open-label, single-arm, Phase I/II trial of human retinal progenitor cells (jCell) for the treatment of retinitis pigmentosa (RP). Study subjects will be screened for eligibility, informed consent obtained, baseline studies of primary and exploratory endpoints performed. Then the subjects will be treated with one of four doses of jCell, with initially enrolled subjects receiving the lowest dose.

### Cohort 1: BCVA no better than 20/200 and no worse than Hand Motions

The first four subjects in Cohort 1 will receive an intravitreal injection of  $0.5 \times 10^6$  hRPC (50  $\mu$ L volume) into the eye with the worst visual acuity; only one eye will be injected. Subjects will be monitored closely following injection for 60 minutes prior to being released home on the day of treatment, based on intraocular pressure <30mm Hg and vital signs returned to pre-injection. Subjects will be treated with ophthalmic corticosteroid eye drops to minimize any inflammation from injection for up to 14 days (including tapering schedule). There will be a minimum four week interval between the

treatment of the first and second subjects in this cohort to confirm no serious injection related AEs have occurred for subject #1 prior to treatment of subject #2. Subsequent cohort 1 subjects at the same dose level will be spaced at least one week apart (subjects 2, 3 and 4). All subjects will receive injection of cells into the eye with the poorest visual acuity. Following at least one week of safety observations for the last study subject at the lower dose level, safety and tolerability data will be reviewed by the DSMB.

Assuming no unexpected safety issues, an additional 4 subjects will be enrolled in Cohort 1 and treated at the second dose level, 1.0 x 10<sup>6</sup> hRPC. Treatment will be similar to the first four subjects, i.e. intravitreal injection under topical anesthesia with treatment of the first two subjects separated by at least 4 weeks and subsequent subjects in this cohort (subject 6, 7 and 8) spaced at least one week apart. Following at least one week of safety observation for the last Cohort 1 subject, safety and tolerability data will be reviewed by the DSMB prior to initiation of Cohort 2.

Following completion of DSMB review of the first 8 subjects in Cohort 1 (dose levels  $0.5 \times 10^6$  and  $1\times 10^6$  hRPC), an additional three subjects may be enrolled into Cohort 1 and treated at the third dose level,  $2\times 10^6$  hRPC ( $50\mu$ L volume). Treatment will be administered as described above for the first two dose levels, with all subjects spaced at least a week apart. Following at least one week of safety observations for the last study subject at the  $2\times 10^6$  hRPC dose level, safety and tolerability data will be reviewed by the DSMB. Assuming no unexpected safety issues and with DSMB recommendation, an additional 3 subjects may be enrolled into Cohort 1 for treatment at the highest dose level,  $3.0\times 10^6$  hRPC ( $50\ \mu$ L volume). Treatment will be administered as described above for the first two dose levels, with all subjects spaced at least a week apart.

### Cohort 2: BCVA no better than 20/40 and no worse than 20/200

The first four subjects in Cohort 2 will receive an intravitreal injection of  $0.5 \times 10^6$  hRPC into the eye with the worst visual acuity; only one eye will be injected. Subjects will be monitored closely following injection for 60 minutes prior to being released home on the day of treatment, based on intraocular pressure <30mm Hg and vital signs returned to pre-injection. Subjects will be treated with ophthalmic corticosteroid eye drops to minimize any inflammation from injection for up to 14 days (including tapering schedule). Assuming no unexpected safety issues in the low dose group, an additional 4 subjects will be enrolled in Cohort 2 and treated at the second dose level,  $1.0 \times 10^6$  hRPC.

Once the first two dose levels are completed in Cohort 2, and following the review of safety data from Cohort 1 subjects who were treated at the third dose level  $(2.0 \times 10^6 \text{ hRPC})$ , three additional subjects may be enrolled into Cohort 2 and treated at the  $2 \times 10^6$ 

hRPC dose level. Following this and assuming no unexpected safety issues in the Cohort 1 subjects at the  $3 \times 10^6$  dose level, three additional subjects may be enrolled into Cohort 2 and treated at this highest dose level.

Assuming safety and tolerability data from all dose levels in Cohort 1 are acceptable, there will be no minimum interval between treatment of subjects in Cohort 2.

If ≥2 subjects develop the same CTCAE grade 3 adverse events or 1 subject develops a CTCAE grade 4 adverse events, the study will be suspended until the DSMB reviews the events and makes a determination whether to continue. If a Grade 3 or worse event is clearly attributable to a non-treatment event and therefore not a suspected adverse reaction, the event will not be considered for the purposes of stopping.

The schedule of observations and assessments during the study are summarized in Table 2 of the study protocol.

#### 4. DETERMINATION OF SAMPLE SIZE

The sample size for this study was not based on any formal statistical considerations.

#### 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using summary tables and listings (TLs). The International Conference on Harmonization (ICH) numbering convention will be used for all TLs. Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories. Percentages for missing values are omitted and do not account for the percent calculation of other categories. Percentages are routinely based on the total category count excluding the missing category if not otherwise mentioned. Percentages showing a rate relative to the total number of subjects in this group are given in special tables (e.g. AE tables). Footnotes will specify the percent basis. All summary tables will be presented by cohort and dose level. Baseline summaries will also include a total summary column. Unless otherwise noted, baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

Individual subject data obtained from the case report forms (CRFs) and derived data will be presented by subject in data listings.

The analyses described in this plan are considered *a priori*, in that they have been defined prior to database lock. Post-hoc analyses will be labeled as such on the output and identified in the CSR.

All analyses and tabulations will be performed using SAS® Version 9.4 or higher. Tables, listings, and figures will be presented in RTF format. Upon completion, all SAS® programs will be validated by an independent programmer. In addition, all program output will undergo a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy, consistency with this plan, consistency within tables, and consistency between tables and corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

#### 6. ANALYSIS POPULATIONS

The following subject population will be used for safety analyses:

• Safety population will include all subjects who received any amount of study drug.

The following subject population will be used for efficacy analyses:

• Intent-to-Treat (ITT) population will include all subjects enrolled and who provide any post-screening data. Subjects in the clinical database will be considered to be enrolled in the study.

# 7. STUDY POPULATION

### 7.1 Subject Disposition

Subject disposition information will be summarized for all subjects by cohort and dose level. Summaries will include: the number of enrolled subjects, the number of subjects in each analysis population, and the primary reason for discontinuation.

### 7.2 Protocol Deviations

Major protocol deviations that could potentially affect the efficacy or safety conclusions of the study will be identified prior to database lock. Major protocol deviations may include, but are not limited to:

- Subjects who did not satisfy selected inclusion and exclusion criteria;
- Subjects who received the incorrect dose;
- Subjects who received an excluded concomitant treatment.

All protocol deviations will be presented in a listing by cohort, dose level and deviation category,

# 7.3 Demographic and Baseline Characteristics

Demographic variables include: age, sex, ethnicity, and race. Age will be calculated in years relative to the informed consent date. Other baseline characteristics include: Medical history, Ocular medical history, height, weight, and study eye (OD [right] or OS [left]).

Descriptive statistics will be presented for age, height, and weight. Frequency counts and percentages will be presented for sex, ethnicity, race, study eye, ocular medical history. Demographic and baseline characteristics will be summarized for the Safety and ITT populations. If safety and ITT populations are identical, the two tables will be combined into a single summary.

Ocular medical history (OMH) will be summarized for each treatment by primary System organ class and dictionary-derived term by using MedDRA 18.1. These summaries will present the number and percentage of subjects per each OMH. Subjects may have more than one OMH per System Organ Class (SOC) and Dictionary Derived Term (DDT). At each level of subject summarization, a subject is counted once if he/she reported one or more OMH at that level. Each summary will be ordered by descending order of incidence of SOC and DDT within each SOC.

Medical history will be presented in a listing.

### 7.4 Prior and Concomitant Medications

Prior and concomitant medication verbatim terms on case report forms (CRFs) will be mapped to Anatomical/Therapeutic/Chemical (ATC) class and Preferred Names using the World Health Organization (WHO) Drug Dictionary Enhanced (version March 1, 2015).

Prior and concomitant medications will be presented in a listing.

#### 8. EFFICACY ANALYSES

The primary efficacy analysis will be based on the ITT population.

# 8.1 Efficacy Variables

The response to jCell injection will be assessed based on the following:

- Best Corrected Visual Acuity (BCVA): BCVA will be measured with the
  electronic visual acuity testing algorithm (E-ETDRS). For each time point
  assessed, the total number of letter missed using E-ETDRS will be recorded for
  each eye and recorded on the Best Corrected Visual Acuity (BCVA) case report
  form.
- Electroretinogram (ERG): For each eye, A-wave Amplitude, B-wave Amplitude, Time from Flash Onset to A-wave Trough and Time from Flash Onset B-wave peak will be measured under the following conditions:
  - o Dark adapted 0.01 ERG (rod response)
  - o Dark adapted 3.0 ERG (rod-cone response)
  - o Light adapted 3.0 ERG (single flash cone response)
  - Light adapted 3.0 flicker ERG

In addition, an overall assessment of Normal or Abnormal will be recorded for each condition. For those assessments of Abnormal, whether the assessment was Clinically Significant will also be reported. If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.

• Optical Coherence Tomography (OCT): for assessment of OCT, the central subfield thickness reported on the Optical Coherence Tomography case report

form will be used. Also information recorded at each visit as to whether Cystoid macular edema (CME) was present and if so, did it involve the foveal center will also be considered.

- Fluorescein Angiography: information regarding active leakage (Yes/No) and ischemia (Yes/No) will be collected for each eye for each Fluorescein Angiography performed.
- Autofluorescence: an overall assessment of Normal or Abnormal will be recorded for each eye for each fundus auto fluorescence imaging performed. For those assessments of Abnormal, whether the assessment was Clinically Significant will also be reported. If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.
- Visual Field Test: an overall assessment of Normal or Abnormal will be recorded for each eye for each visual field examination performed. For those assessments of Abnormal, whether the assessment was Clinically Significant will also be reported. In addition, information regarding Mean Deviation, Fixation Loss, False Positives and False Negatives will also be recorded. If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.

# 8.2 Baseline Values

Unless otherwise noted, baseline is defined as the value obtained at baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

# 8.3 Handling of Dropouts or Missing Data

No imputations will be made for missing values. Summaries will be based on observed data only.

# 8.4 Interim Analysis and Data Monitoring

There are no planned interim analyses for this study.

# 8.5 Examination of Subgroups

There are no planned subgroup analyses for this study.

# 8.6 Multiple Comparison/Multiplicity

No adjustments for multiplicity will be made in this study.

#### 8.7 Multicenter Studies

Analyses to compare differences in response by center or any treatment by center interactions are not planned.

#### 9. METHODS OF EFFICACY ANALYSIS

Since this is an exploratory study, no formal hypothesis testing will be done. Descriptive statistics will be used to tabulate and summarize study outcomes. The baseline results of clinical examinations of the non-injected (non-study) eye serve as controls for the injected (study) eye. Results of clinical testing of the non-injected eye will also be described. Continuous variables will be summarized descriptively (sample size, mean, standard deviation and error, minimum and maximum). Discrete variables will be summarized by frequency or percentage. All efficacy analyses will be based on the ITT Population. All efficacy variables will be presented by cohort and dose level using summary statistics.

# 9.1 Best Corrected Visual Acuity (BCVA)

For BCVA, summary statistics of the total number of letters correct (Letters correct=100-letters missed) will be generated at each time point for each cohort. Separate tables will be created for the Study Eye and the Non-Study Eye. In addition, change from baseline will also be summarized for each post baseline time point. For individual subjects who have number scores, the same formula for letters correct will be used to calculate each time point (letters correct = 100-letters missed). For subjects who do not have a number score e.g. counting fingers (CF), hand motions (HM) or no light perception )NLP), letters missed will be considered to be 100 and letters correct will therefore be zero. summarized (i) proportion of treated eyes with  $\geq$ 5,  $\geq$ 10 and  $\geq$ 15 letter

improvements at any timepoint in the study same for untreated eyes at month 3,6,9 and 12 or Early Termination.

In addition, change in BCVA from baseline will be summarized for each dose level combining cohorts 1 and 2 at month 3,6,9 and 12 or early termination. Difference of mean change in BCVA between treated eye and non-treated eye from baseline will be summarized at month 3,6,9 and 12 or early termination. Furthermore, proportion of  $\geq$ 5,  $\geq$ 10 and  $\geq$ 15 letter improvements will be summarized for each dose level combining cohorts 1 and 2 at month 3,6,9 and 12 or early termination.

# 9.2 Electroretinogram (ERG)

Electroretinogram (ERG) results will be summarized using both continuous and categorical methods. Descriptive statistics by eye (Study, Non-Study) of A-wave Amplitude, B-wave Amplitude, Time from Flash Onset to A-wave Trough and Time from Flash Onset B-wave peak endpoints will be calculated for each time point and condition specified in Section 8.1. Summaries of change from baseline will be presented in a similar fashion. In addition, count and percentages of overall ERG assessments of the following categories will be shown for each time point, eye (Study, Non-Study) and condition specified in Section 8.1:

- Normal
- Abnormal, Not Clinically Significant (NCS)
- Abnormal, Clinically Significant (CS)

#### 9.3 Visual Field Examination

From the visual field examination, whether the results are Normal, Abnormal NCS and Abnormal CS will be summarized with counts and percentages at each time point for both study eye and non- study eye.

#### 10. SAFETY ANALYSES

All safety analyses will be based on the Safety population. Adverse events will be monitored by the investigator and the subject. The safety analyses of laboratory parameters will include descriptive statistics and AEs will include frequency counts and percentages. Summaries of AEs will be generated by type (AE or SAE), body system and preferred term, severity, and relationship to study product.

# 10.1 Study Drug Administration

Treatment compliance will be assessed via direct observation by the study investigator who is responsible for study drug administration. The cell dose and exact time of injection will be recorded. Study drug administration responses will be tabulated for each treatment according to questions asked in the CRF, including whether the total dose was administered, whether there were any dose interruptions were there any AEs observed, were the subject's vital signs comparable to pre-treatment of study drug injection, was the subject's IOP measurement less than 30 mm post treatment of study drug injection and was the subject prescribed topical treatment after treatment of study drug injection.

#### 10.2 Adverse Events

All adverse event summaries will be restricted to Treatment Emergent Adverse Events (TEAE), which are defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. If it cannot be determined whether the AE is treatment emergent due to a partial onset date then it will be counted as such. Verbatim terms on case report forms will be mapped to preferred terms and system organ classes using the Medical Dictionary for Regulatory Activities (MedDRA) (version 18.1).

Each adverse event summary will be displayed by treatment group. Summaries that are displayed by system organ class and preferred terms will be ordered by descending order of incidence of system organ class and preferred term within each system organ class. Summaries of the following types will be presented:

- Subject and event incidence of TEAEs by MedDRA system organ class and preferred term.
- Subject incidence of TEAEs by MedDRA system organ class, preferred term, and highest severity. At each level of subject summarization a subject is classified according to the highest severity if the subject reported one or more events. Categories of severity will be "Mild", "Moderate", "Severe" and "Life Threatening" in this summary. The "Life Threatening" column will only be shown if at least 1 life-threatening AE is reported. If any AEs are reported with missing severity, then a footnote will be added to indicate how many AEs with missing severity were reported.
- Subject and event incidence of related TEAEs by MedDRA system organ class and preferred term. Related AEs are those reported as "Related", "Possibly Related" or relationship was not reported. At each level of subject summarization a subject is classified according to the closest relationship if the subject reported

- one or more events. AEs with a missing relationship will be considered related for this summary.
- Subject and event incidence of serious TEAEs by MedDRA system organ class and preferred term.

# 10.3 Clinical Laboratory Evaluation

Hematology, serum chemistry and coagulation laboratory parameters will be summarized using descriptive statistics at baseline, Day 7, Day 28, Month 3, Month 6, and Month 12/Early Term. Change from baseline in the laboratory parameters will also be presented, Unless otherwise noted, baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

No concerns are expected regarding the drug for laboratory results since the drug is expected to stay in the eye. As a result, no analysis using high/low flags will be carried out.

Urinalysis results will not be summarized but will be provided in data listing. Separate listing of abnormal clinically significant lab values and ECG interpretation will be presented.

# 10.4 Vital Signs

Vital signs (systolic BP, diastolic BP, heart rate, respiration, temperature, and weight) will be summarized using descriptive statistics at baseline and at each post-baseline time point. Changes from baseline will also be summarized. Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

# 10.5 Physical Examination

Physical examination results will be included in data listings only.

### 10.6 Electrocardiogram

ECG parameters will be presented in a listing..

# 10.7 Ophthalmic AEs

# 10.7.1 Slit Lamp and Fundus Photography

Slit Lamp and Fundus Photography - The slit lamp exam will be summarized by eye structure. For eye structures of eyelids, eyelashes, conjunctiva, sclera, cornea, and iris, subjects will be tabulated by the categories of Normal, Abnormal NCS, and Abnormal CS at each time point, and percentages will be displayed. For anterior chamber flare, subjects will be tabulated by the flare grade and the categories of Abnormal NCS and Abnormal CS. For lens status, subjects will be tabulated as aphakic, pseudophakic, and phakic. For cataract type, subjects will be tabulated as nuclear, cortical, posterior sub capsular, and not applicable. Subjects will also be tabulated by grades of 1+, 2+, 3+ and 4+. For the fundus photography, subjects will be tabulated by the categories of Normal and Abnormal NCS and Abnormal CS. Results will be presented for each of subjects' eyes (study eye and non-study eye) at all time points.

If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.

# 10.7.2 Intraocular Pressure (IOP)

IOP - Intraocular pressure and change in intraocular pressure will be summarized descriptively by time point.

#### 10.7.3 B-scan

B-scan results will be tabulated by Normal and Abnormal results at each time point and overall results will be counted as good or poor. B-scan results will also be tabulated by whether injected cells were visualized. If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.

# 10.7.4 Dilated Fundoscopic Examination

Dilated Fundoscopic Examination- for the vitreous exam, optic nerve exam, macula exam, and peripheral retina exam, counts and percentages of Normal, Abnormal NCS and Abnormal CS will be presented by eye and time point. When available, summaries of Severity (Mild +1, Moderate +2, Severe +3, Very Severe +4) will also be included. If Clinically Significant value is not reported in the follow-up visit, then the value will be imputed based on the value of previous visit, consistent with CRF completion guidelines. For example, if abnormal change from previous visit is "NO" then imputed value will be value from the previous visit.

# 10.7.5 Post Injection Clinical Vitreous Exam

Post Injection Clinical Vitreous Exam, counts and percentages will be summarized for method used (indirect ophthalmoscopy, fundus exam, slit lamp exam and other) and observations (cells, clumps, opacity, debris, strands, inflammation and other).

# 10.7.6 Optical Coherence Tomography (OCT)

OCT results will be summarized in a table showing the counts and percentages of subjects whose eyes (both study eye and non-study eye) show cystoid macular edema present, and of those who do, how many cases involve the foveal center.

# 10.7.7 Fluorescein Angiography

For fluorescein angiography analysis, the number of subjects whose eyes (both study and non-study eye) have active leakage or show signs of ischemia at each time point will be shown by frequency and corresponding percentages.

#### 10.7.8 Autofluorescence

Fundus auto fluorescence will be summarized for both study eye and non-study eye at each time point with counts and incidence rates for each of the possible options of Normal, Abnormal NCS, Abnormal CS

#### 11. REFERENCES

 $\underline{http://www.rand.org/content/dam/rand/www/external/health/surveys\_tools/vfq/vfq25\_ma\_nual.pdf}$ 

Mangione, CM, Lee PP, Gutierrez, PR, et al. Development of the 25-item National Eye Institute Visual Function Questionnaire (VFQ-25). Archives of Ophthalmology, 2001. 119: 1050-1058.

http://eva.jaeb.org/test\_information/Algorithm\_EETDRS.pdf

### **APPENDICES**

# **Appendix A: Presentation of Data and Programming Specifications**

#### General

- Specialized text styles, such as bold, italics, borders, shading, superscripted and subscripted text will not be used in tables and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters are to be used in tables and data listings.
- Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used on a table or data listing.
- Hexadecimal character representations are allowed (e.g.,  $\mu$ , a,  $\beta$ ).
- All footnotes will be left justified and at the bottom of a page. Footnotes should be used sparingly and must add value to the table or data listing.

#### **Tables**

- Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.
- Means and medians will be presented to one more decimal place than the raw data. Standard deviations will be presented to two more decimal places than the raw data. Minimums and maximums will be reported with the same number of decimal places as the raw data.
- Percentages will be presented to the tenths place.
- For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up," this reason will be included in the table with a count of 0. Categories with zero counts will not have zero percentages displayed.

#### Listings

- Formal organization of the listing may be changed during programming if appropriate, e.g., additional variables may be included, change in the column order, or the listing may be split into multiple parts due to space constraints, etc.
- If not otherwise specified, all data listings will be sorted by sequence/treatment, center, subject number, visit, and date/time as appropriate.
- All date values will be presented in a SAS date (e.g., 29AUG2001) format.

• All observed time values will be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds will only be reported if they were measured as part of the study.

# Missing or incomplete dates (i.e., AEs and concomitant medications)

The most conservative approach will be systematically considered. If the AE onset date is missing / incomplete, it is assumed to have occurred during the study treatment phase (i.e., considered a TEAE) except if the partial onset date or other data such as the stop date, indicates differently. Similarly, a medication with partial start and stop dates could be considered as both a prior and concomitant treatment.

The following algorithms will be applied to missing and incomplete start and stop dates:

### **Start Dates**

- If the day portion of the start date is missing, then the start date will be estimated to be equal to the date of first dose of study drug, provided the start month and year are the same as the first dose of study drug and the stop date is either after the first dose of study drug or completely missing. Otherwise, the missing day portion will be estimated as '01'.
- If both the day and month portions of the start date are missing, then the start date will be estimated to be equal to the date of first dose of study drug, provided the start year is the same as the first dose of study drug and the stop date is either after the first dose of study drug or completely missing. Otherwise, the event will be assumed to start on the first day of the given year (e.g., ??-???-2013 is estimated as 01-JAN-2013).
- If the start date is completely missing and the stop date is either after the dose of study drug or completely missing, the start date will be estimated to be the day of study drug dosing. Otherwise, the start date will be estimated to be the first day of the same year as the stop date. All other non-AE and non-concomitant medication day calculations where only partial dates are available will be handled as follows: the first day of the month will be used in the calculations if the day part of a start date is missing while January 1 will be employed if both the month and day parts of a start date are missing.

#### **Stop Dates**

• If only the day of resolution is unknown, the day will be assumed to the last of the month (e.g., ??-JAN-2013 will be treated as 31-JAN-2013).

- If both the day and month of resolution are unknown, the event will be assumed to have ceased on the last day of the year (e.g., ??-???-2013 will be treated as 31-DEC-2013).
- If the stop date is completely missing or the event is continuing, the event will be assumed to be after first dose of study drug and will be imputed using the last known date on the study.

# Appendix B: List of Tables, Figures, and Listings

The following TLF numbering is completed according to ICH guidelines. The ICH heading number and description are in **bold**. Minor changes from this planned index do not need to be amended in the SAP.

Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.

# **List of Tables**

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| 14.1 | | DEMOGRAPHIC DATA |
| | 14.1.1 | Subject Disposition |
| | 14.1.2 | Demographic and Baseline Characteristics (Safety/ITT |
| | | Population) |
| | 14.1.3 | Ocular Medical History at Baseline (Safety/ITT Population) |
| 14.2 | | EFFICACY DATA |
| | 14.2.1.1 | Best Corrected Visual Acuity (ETDRS): Study Eye |
| | 14.2.1.2 | Best Corrected Visual Acuity (ETDRS): Non-Study Eye |
| | 14.2.1.3 | Categorical Analysis of Best Corrected Visual Acuity |
| | | (ETDRS): Study Eye |
| | 14.2.1.4 | Categorical Analysis of Best Corrected Visual Acuity |
| | | (ETDRS): Non-Study Eye |
| | 14.2.1.5 | Best Corrected Visual Acuity (ETDRS): by Dose Level |
| | | Study Eye Vs Non-Study Eye |
| | 14.2.1.6 | Categorical Analysis of Best Corrected Visual Acuity |
| | | (ETDRS): by Dose Level Study Eye Vs Non-Study Eye |
| | 14.2.2.1 | Electroretinogram (ERG), Categorical Analysis: Study Eye |
| | | (ITT Population) |
| | 14.2.2.2 | Electroretinogram (ERG), Categorical Analysis: Non-Study |
| | | Eye (ITT Population) |
| | 14.2.3 | Visual Field Examination by Eye, Categorical Analysis (ITT |
| | | Population) |
| 14.3 | | SAFETY DATA |
| | 14.3.1 | Study Drug Administration (Safety Population) |
| 14.3.1 | | Displays of Adverse Events |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| | 14.3.1.1 | TEAEs by System Organ Class and Preferred Term (Safety |
| | | Population) |
| | 14.3.1.2 | TEAEs by System Organ Class, Preferred Term and |
| | | Maximum Severity (Safety Population) |
| | 14.3.1.3 | Related to Study Drug TEAEs by System Organ Class and |
| | | Preferred Term (Safety Population) |
| | 14.3.1.4 | Serious TEAEs by System Organ Class and Preferred Term |
| | | (Safety Population) |
| | 14.3.4.1 | Hematology (Safety Population) |
| | 14.3.4.2 | Chemistry (Safety Population) |
| | 14.3.4.3 | Coagulation (Safety Population) |
| | 14.3.4.4 | Vital Signs (Safety Population) |
| | 14.3.4.5 | 12-Lead Electrocardiogram-Overall Interpretation (Safety |
| | | Population) |
| | 14.3.4.6.1 | Slit Lamp Examination: Study Eye (Safety Population) |
| | 14.3.4.6.2 | Slit Lamp Examination: Non-Study Eye (Safety Population |
| | 14.3.4.7 | Fundus Photography by Eye (Safety Population) |
| | 14.3.4.8.1 | Intraocular Pressure (IOP): Study Eye (Safety Population) |
| | 14.3.4.8.2 | Intraocular Pressure (IOP): Non-Study Eye (Safety |
| | | Population) |
| | 14.3.4.9.1 | B-Scan: Study Eye (Safety Population) |
| | 14.3.4.9.2 | B-Scan: Non-Study Eye (Safety Population) |
| | 14.3.4.10.1 | Dilated Fundoscopic Examination: Study Eye (Safety |
| | | Population) |
| | 14.3.4.10.2 | Dilated Fundoscopic Examination: Non-Study Eye (Safety |
| | | Population) |
| | 14.3.4.11 | Post Injection Clinical Vitreous Exam: Study Eye (Safety |
| | | Population) |
| | 14.3.4.12.1 | Optical Coherence Tomography (OCT): Study Eye, |
| | | Categorical Analysis (ITT Population) |
| | 14.3.4.12.2 | Optical Coherence Tomography (OCT): Non-Study Eye, |
| | | Categorical Analysis (ITT Population) |
| 14.3 | 14.3.4.13.1 | Fluorescein Angiography: Study Eye, Categorical Analysis (ITT Population) |
| | 14.3.4.13.2 | Fluorescein Angiography: Non-Study Eye, Categorical Analysis (ITT Population) |

jCyte, Inc. Statistical Analysis Plan
Protocol: JC-01 08Nov2017

| ICH | Table | |
|---------|-------------|--------------------------------------------------|
| Heading | Number | Table Description |
| | 14.3.4.14.2 | Autofluorescence: Non-Study Eye (ITT Population) |

# **List of Data Listings**

| ICH | Listing | |
|---------|-------------|--------------------------------------------------|
| Heading | Number | Listing Description |
| 16.2.1 | 16.2.1.1 | Subject Disposition |
| 16.2.2 | 16.2.2.1 | Protocol Deviations |
| | 16.2.2.2 | Inclusion/Exclusion Criteria |
| 16.2.4 | 16.2.4.1 | Demographics and Baseline Characteristics |
| | 16.2.4.2 | Medical History |
| | 16.2.4.3 | Ocular Medical History |
| | 16.2.4.4 | Urine Drug Screen |
| | 16.2.4.5 | Infectious Disease Tests |
| 16.2.5 | 16.2.5 | Study Drug Administration |
| 16.2.6 | 16.2.6.1 | Best Corrected Visual Acuity (ETDRS) |
| | 16.2.6.2 | Electroretinogram |
| | 16.2.6.3 | Optical Coherence Tomography (OCT) |
| | 16.2.6.4 | Fluorescein Angiography |
| | 16.2.6.5 | Autofluorescence |
| | 16.2.6.6 | Visual Field Examination |
| 16.2.7 | 16.2.7.1 | Adverse Events |
| | 16.2.7.2 | Serious Adverse Events |
| | 16.2.7.3 | Related Adverse Events |
| | 16.2.7.4 | Post Injection Clinical Vitreous Exam |
| 16.2.8 | 16.2.8.1 | Hematology |
| | 16.2.8.2 | Chemistry |
| | 16.2.8.3 | Coagulation |
| | 16.2.8.4 | Urinalysis |
| | 16.2.8.5 | Clinically Significant Lab Values |
| | 16.2.8.6 | Vital Signs |
| | 16.2.8.7.1 | 12-Lead Electrocardiogram |
| | 16.2.8.7.2 | Clinically Significant 12-Lead Electrocardiogram |
| | | Interpretation |
| | 16.2.8.8 | Physical Examination |
| | 16.2.8.9 | Prior and Concomitant Medications |
| | 16.2.8.10 | Pregnancy Test |
| | 16.2.8.11 | PRA and DRA Antibody Test Results Received |
| | 16.2.8.12 | HLA Antibody Testing |
| | 16.2.8.13 | RP Gene Mutation Recieved |
| | 16.2.8.14.1 | Slit Lamp (OS) |

| ICH | Listing | |
|---------|-------------|---------------------------------|
| Heading | Number | Listing Description |
| | 16.2.8.14.2 | Slit Lamp (OD) |
| | 16.2.8.15 | Fundus Photography |
| | 16.2.8.16 | Intraocular Pressure (IOP) |
| | 16.2.8.17 | B-Scan |
| | 16.2.8.18 | Dilated Fundoscopic Examination |

**Appendix C: Table Layouts** 

Protocol: JC-01

**Table 14.1.1 Subject Disposition** All Enrolled Subjects

| | | Coh | ort 1 | | | Coh | ort 2 | | |
|---|---|---|---|---|---|---|---|---|---|
| | $0.5 \times 10^6$ | 1.0 x 10 <sup>6</sup> | $2.0 \times 10^6$ | $3.0 \times 10^6$ | $0.5 \times 10^6$ | 1.0 x 10 <sup>6</sup> | $2.0 \times 10^6$ | $3.0 \times 10^6$ | |
| | hRPC | hRPC | hRPC | hRPC | hRPC | hRPC | hRPC | hRPC | Total [1] |
| Subjects Enrolled | N | N | N | N | N | N | N | N | N |
| ITT Population [2] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Safety Population [3] | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Primary Reason for Discontinuation | | | | | | | | | |
| Completed Study | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Adverse Event | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Lack of Efficacy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Lost to Follow Up | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Non-Compliance with Study Treatment | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Physician Decision | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Pregnancy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Progressive Disease | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Protocol Deviation | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Recovery | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Study Terminated by Sponsor | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Withdrawn by Subject | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Death | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t program.sas date time

Programmer Note: only shows primary reason for Discontinuation that has results.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] All enrolled subjects who provide any post-screening data.
[3] Received any amount of jCyte treatment.
Note: Percentages based on Subjects Enrolled.

**Table 14.1.2 Demographic and Baseline Characteristics** Safety/ITT Population

| | Cohort 1 | | | | Cohort 2 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | $0.5 \times 10^6$ | $1.0 \times 10^6$ | $2.0 \times 10^6$ | $3.0 \times 10^6$ | $0.5 \times 10^6$ | 1.0 x 10 <sup>6</sup> | $2.0 \times 10^{6}$ | $3.0 \times 10^6$ | Total [1] |
| | hRPC | hRPC | hRPC | hRPC<br>(N=) | hRPC | hRPC | hRPC<br>(N=) | hRPC | (N=) |
| | (N=) | (N=) | (N=) | | (N=) | (N=) | | (N=) | |
| Age (years) [2] | | | | | | | | | |
| n | n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Sex | (0/) | (0/) | (0/) | (0/) | (0/) | (0./) | (0/) | (0./) | (0/) |
| Male | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ethnicity | | | | | | | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Race | | | | | | | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Multiple Races Checked | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ' 1 1 1 4 C 1 4 1 12 | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |

Total includes both Cohorts 1 and 2.

[2] Age determined by comparing date of birth to date of informed consent.

[3] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

**Table 14.1.2 Demographics and Baseline Characteristics** Safety/ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | •••• | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | •••• | Total <sup>[1]</sup><br>(N=) |
| Study Eye | | | | | |
| OD (Right) | n (%) | n (%) | n (%) | n (%) | n (%) |
| OS (Left) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Height (cm) [3] | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Weight (kg) [3] | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |

Programmer note: For the subsequent tables, use Table 14.1.2 to determine which columns to include.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] Age determined by comparing date of birth to date of informed consent.
[3] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date time

**Table 14.1.3** Ocular Medical History Safety/ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| Ocular System Organ Class//<br>Dictionary Derived Term | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup> (N=) |
| Congenital, Familial and Genetic Disorders<br>Dictionary Derived Term | | | | | |
| Eye Disorders<br>Dictionary Derived Term | n (%) | n (%) | n (%) | n (%) | n (%) |
| Nervous System Disorders<br>Dictionary Derived Term | n (%) | n (%) | n (%) | n (%) | n (%) |
| Surgical Medical Procedures Dictionary Derived Term | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2. path\t\_program.sas date time

Programmer Note: add all SOC and PT terms from xmh1 dataset.. Programmer Note:sort table by Alphabetical SOC order.

Table 14.2.1.1
Best Corrected Visual Acuity (ETDRS): Study Eye
Number of Letters correct
ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup><br>(N=) |
| Baseline [2] | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | xx.x | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1 | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX.X | xx.x | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1 Change from Baseline | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |
| Day 2 | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | ••• | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Day 3, Day 7, Day14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12 or Early Term. Programmer Note: Table 14.2.1.2 will contain the same information for the Non-Study Eye

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time
**Table 14.2.1.3** Categorical Analysis of Best Corrected Visual Acuity (ETDRS): Study Eye **Number of Letters correct ITT Population** 

| | Cohort | 1 | Cohor | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | $0.5 \times 10^{6} hRPC$ | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Proportion of Subjects with Specified increase in letters correct for any Post | (n=) | (n=) | (n=) | (n=) | (n=) |
| Baseline Assessment | | , , | | . , | ` / |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 3 | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 9 | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 12 or | (n=) | (n=) | (n=) | (n=) | (n=) |
| Eartly Termination | | | | | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) |

[1] Total includes both Cohorts 1 and 2. path\t\_program.sas date

Programmer Note: Table 14.2.1.4 will contain the same information for the Non-Study Eye
Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

jCyte, Inc.
Protocol: JC-01

Table 14.2.1.5
Best Corrected Visual Acuity (ETDRS): Study Eye vs Non-Study Eye
Number of Letters correct
ITT Population

| | $0.5 \times 10^6 hRPC$ | | 1.0 x | 10 <sup>6</sup> hRPC | 2.0 x | 10 <sup>6</sup> hRPC | $3.0 \times 10^6 hRPC$ | |
|---|---|---|---|---|---|---|---|---|
| | Study Eye<br>(N=) | Non-Study Eye<br>(N=) | Study Eye<br>(N=) | Non-Study Eye<br>(N=) | Study Eye<br>(N=) | Non-Study Eye<br>(N=) | Study Eye<br>(N=) | Non-Study Eye<br>(N=) |
| Baseline [1] | | | | | | | | |
| n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| Month 3 | | | | | | | | |
| n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | xx.x | xx.x | xx.x | XX.X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Month 3 Change from Baseline | | | | | | | | |
| n | n | n | n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X | XX.X | XX.X | xx.x | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Difference between Study Eye Vs Non-Study Eye | | | | | | | | |
| n | | n | | n | | n | | n |
| Mean (SD) | | xx.x (xx.x) | | xx.x(xx.x) | | xx.x (xx.x) | | xx.x (xx.x) |
| Median | | XX.X | | XX.X | | XX.X | | XX.X |
| Min, Max | | xx, xx | | xx, xx | | xx, xx | | xx, xx |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Programmer Note: Continue table for Visits: Month 3, Month 6, Month 9, Month 12 or Early Term.

**Table 14.2.1.6** Categorical Analysis of Best Corrected Visual Acuity (ETDRS): Study Eye vs Non-Study Eye **Number of Letters correct ITT Population** 

| | 0.5 x 1 | 0 <sup>6</sup> hRPC | 1.0 x 1 | 0 <sup>6</sup> hRPC | 2.0 x 10 | <sup>6</sup> hRPC | 3.0 x 10 | ) <sup>6</sup> hRPC |
|---|---|---|---|---|---|---|---|---|
| | Study Eye<br>(N=) | Non-Study<br>Eye (N=) | Study Eye<br>(N=) | Non-Study<br>Eye (N=) | Study Eye<br>(N=) | Non-Study<br>Eye (N=) | Study Eye<br>(N=) | Non-Study<br>Eye (N=) |
| Proportion of Subjects with Specified increase in letters correct for any Post<br>Baseline Assessment | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 3 | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 9 | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Proportion of Subjects with Specified increase in letters correct at Month 12 or Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) | (n=) |
| >=5 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=10 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| >=15 Letters Increase | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t program.sas date time

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point..

**Table 14.2.2.1** Electroretinogram (ERG) - Study Eye **Categorical Analysis** ITT Population

| | Cohor | t 1 | Cohort | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Dark Adapted 0.01 ERG (rod response) | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 12/ Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dark Adapted 3.0 ERG (rod-cone response) | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 12/ Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

Programmer Note: Continue table for Light Adapted 3.0 ERG (single flash cone response), Light Adapted 3.0 Flicker ERG

Total includes both Cohorts 1 and 2.

[2] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date time

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.. Programmer Note: Table 14.2.2.2 will contain the same information for the Non-Study Eye.

**Table 14.2.3** Visual Field Examination by Eye Categorical Analysis
ITT Population

| | Cohor | t 1 | Cohort | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | Total [1] | |
| | (N=) | | (N=) | | (N=) |
| Study Eye | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 12/Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Non-Study Eye | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 12/Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date

| Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point | |
|---|---|
| | Page 43/120 |

Table 14.3.1 Study Drug Administration Safety Population

| | Cohor | t 1 | Cohort | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Eye Drug Injected into: | | | | | |
| OD (Right) | n (%) | n (%) | n (%) | n (%) | n (%) |
| OS (Left) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Total Dose Administered? | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| 110 | 11 (73) | 11 (70) | 11 (70) | 11 (70) | 11 (70) |
| Any Dose interruptions? | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Were any Adverse Events observed? | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subject Vital Signs comparable to pre injection levels? | (0/) | (0/) | (0/) | (0/) | (0/) |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subject IOP < 30mm post treatment of injection? | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| | ( ) | \ <i>\</i> | ( ) | ( ) | ( -) |
| Subject Prescribed Topical Treatment after Study Drug | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| des both Cohorts 1 and 2. | | | | | |

[1] Total includes both Cohorts 1 and 2. path\t\_program.sas date time

**Table 14.3.1.1 TEAEs by System Organ Class and Preferred Term Safety Population** 

| System Organ Class / | 0.5 x 10 | <sup>6</sup> hRPC | | | 0.5 x 10 <sup>6</sup> | hRPC | | | Total <sup>[1]</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | (N=) | | (N=) | | (N= | =) | (N=) | | (N | [=) |
| | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One TEAE | n (%) | xx | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | xx |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| ••• | | | | | | | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once. path\t\_program.sas date time

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

jCyte, Inc. Protocol: JC-01

**Table 14.3.1.2** TEAEs by System Organ Class, Preferred Term and Maximum Severity **Safety Population** 

Cohort 1

| | | 0.5 | x 10 <sup>6</sup> hRPC | | 1011 1 | 1 | | |
|---|---|---|---|---|---|---|---|---|
| System Organ Class / | | 0.3 | (N=) | • | | | | |
| Preferred Term | Mild | Moderate | Severe | Life Threatening | Mild | Moderate | Severe | Life Threatening |
| Subjects Reporting at Least One TEAE | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| • | | | | | | | | |
| · | | | | | | | | |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using maximum severity grade. path\t program.sas date

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

**Table 14.3.1.2** TEAEs by System Organ Class, Preferred Term and Maximum Severity **Safety Population** 

Cohort 2

| | | | | Collo | It Z | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | | | | | | Total [1] | | | |
| System Organ Class / | | | | | | | | | | (N= | = ) | |
| Preferred Term | Mild | Moderate | Severe | Life | Mild | Moderate | Severe | Life | Mild | Moderate | Severe | Life |
| | | | | Threatening | | <del>.</del> | | Threatening | | _ | | Threatening |
| Subjects Reporting at Least One TEAE | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| • | | | | | | | | | | | | |
| · | | | | | | | | | | | | |
| System Organ Class 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 1 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term 2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using maximum severity grade. path\t program.sas date time

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.


**Table 14.3.1.3** Related to Study Drug TEAEs by System Organ Class and Preferred Term Safety Population

| System Organ Class / | 0.5 x 10 | 6 hRPC | | | $0.5 \times 10^6$ | hRPC | | | Total [1] | |
|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | (N=) | | (N=) | | (N= | =) | (N=) | | (N=) | |
| | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One Related TEAE | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | xx |
| System Organ Class 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| ••• | | | | | | | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the closest relationship to study drug. Note: Related Iincludes all events reported as "Possibly Related", "Related" or have missing relationship to study drug. path\t program.sas date time

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

**Table 14.3.1.4** Serious TEAEs by System Organ Class and Preferred Term Safety Population

| System Organ Class / | 0.5 x 10 | 6 hRPC | | | $0.5 \times 10^6$ | hRPC | | | Total [1] | |
|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | (N=) | | (N=) | | (N= | =) | (N=) | | (N=) | |
| | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One Serious TEAE | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | xx |
| System Organ Class 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX | n (%) | XX |
| ••• | | | | | | | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one serious adverse event are counted only once. path\t\_program.sas date

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

Table 14.3.4.1 Hematology Safety Population

| | | Cohort 1 | | Coho | rt 2 | |
|---|---|---|---|---|---|---|
| Laboratory Parameter | Time Point | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | ••••• | Total <sup>[1]</sup><br>(N=) |
| | P 1: [2] | | | | | |
| Hemoglobin (g/dL), | Baseline [2] | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) | xx.x(xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Day 7 | | | | | |
| | Ň | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| | Day 7 Change from Baseline | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | | | | | |
| | Willi, Wax | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | Day 28 | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Day 28, Month 3, Month 6, Month 12/Early Term.

Programmer Note: Table will include the following hematology parameters: Hemoglobin (g/dL), Hematocrit (%), Platelet Count(x 10^3/uL), Red cell Count (x 10^6/uL), White cell Count(x 10^3/uL), Percent Neutrophil(%)s, Percent Lymphocytes(%)s, Percent Monocyte(%), Percent Eosinophil(%), Percent Basophils(%), Neutrophil(x 10^3/uL)s, Lymphocytes(x 10^3/uL), Eosionophil(x 10^3/uL) and Basophils(x 10^3/uL).

<sup>[2]</sup> Baseline is defined as the last non-missing value prior to first dose of study drug. path\t\_program.sas date time

Table 14.3.4.2 Chemistry Safety Population

| | | Cohort 1 | | Coho | Cohort 2 | |
|---|---|---|---|---|---|---|
| | | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| Laboratory Parameter | Time Point | (N=) | | (N=) | | (N=) |
| ALT (SGPT) (U/L) | Baseline [2] | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x(xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| | Day 7 | | | | | |
| | Ň | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX | xx, xx | xx, xx |
| | Day 7 Change from Baseline | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Day 28 | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Day 28, Month 3, Month 6, Month 12/Early Term.

Programmer Note: Table will include the following serum chemistry parameters: ALT (SGPT) (U/L), AST (SGOT) (U/L), Alkaline Phosphatase (U/L), Bilirubin (mg/dL), Sodium (mmol/L), Potassium (mmol/L), Chloride (mmol/L), Bicarbonate (mmol/L), Blood Urea Nitrogen (mgdL), Creatinine (mg/dL), Total Protein (g/dL), Albumin (g/dL), Calcium(mg/dL), Phosphate (mg/dL) and Glucose (mg/dL).

Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

**Table 14.3.4.3** Coagulation **Safety Population** 

| | | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|---|
| | | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| Laboratory Parameter | Time Point | (N=) | | (N=) | | (N=) |
| Prothrombin Time (PT) | Sec) Baseline [2] | | | | | |
| roundinam rime (r r) ( | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Day 7 | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Day 7 Change from Baseline | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Day 28 | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | xx.x | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | ••• | ••• | | | | ••• |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Day 28, Month 3, Month 6, Month 12/Early Term.

Programmer Note: Table will include the following Coagulation parameters: Partial Thromboplastin Time (PTT) (sec) and INR.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date

**Table 14.3.4.4 Vital Signs Safety Population** 

| | | Coho | ort 1 | Coho | Cohort 2 | |
|---|---|---|---|---|---|---|
| Vital Sign | Time Point | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | ••••• | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup><br>(N=) |
| Systolic BP (mmHg) | Baseline [2] | | | | | |
| bystone Dr (mining) | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | iviiii, iviax | AA, AA | AA, AA | AA, AA | AA, AA | AA, AA |
| | Day 0 15 min Post-Injection | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Day 0 15 min Post-Injection | | | | | |
| | Change from Baseline | | | | | |
| | N | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| | ivini, iviax | лл, лл | лл, лл | лл, лл | лл, лл | лл, лл |
| | Day 2 | | | | | |
| | n | n | n | n | n | n |
| | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | XX, XX | xx, xx | XX, XX | XX, XX | XX, XX |
| | • | • | * | , | • | |
| | | ••• | ••• | | ••• | |

Source: xxx

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

Programmer Note: Table will include the following vital signs: systolic BP (mmHg), diastolic BP (mmHg), Heart Rate (bpm), Respiration (Breaths/min) and Temperature(C).

| Programmer Note: Continue table for Visits: Day 0-60 min post injection, Day 1, Day 2, Day 3, Day 7, Day 14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term. | |
|---|---|
| Paį | ge 54/1 |

jCyte, Inc. Protocol: JC-01 Page 1 of x

**Table 14.3.4.5** 12-Lead Electrocardiogram – Overall Interpretation Safety Population

| | Cohor | Cohort 1 | | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup><br>(N=) |
| Baseline [2] | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 1 | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that Perticular time point.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

**Table 14.3.4.6.1** Slit Lamp Examination: Study Eye **Safety Population** 

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Eyelids | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 2 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 3 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 7 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

ath\t program.sas date

Programmer Note: Continue table for Eyelashes, Conjunctiva, Sclera, Cornea, Anterior Chamber Flare), Iris, Lens Status, Cataract Type, Grade.

Programmer Note: Continue table for Visits: Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term.

Programmer Note: Table 14.3.4.6.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that Perticular time point..

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

<sup>[3]</sup> Subject may be counted more than one row.

Programmer Note: Table can be modified to align with information collected on the CRF.

Table 14.3.4.6.1 Slit Lamp Examination: Study Eye **Safety Population** 

| | Cohort | Cohort 1 | | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Lens Status | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Aphakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Psedophakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Phakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Aphakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Psedophakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Phakic | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cataract Type [3] | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Nuclear | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cortical | n (%) | n (%) | n (%) | n (%) | n (%) |
| Posterior Subcapsular | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Nuclear | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cortical | n (%) | n (%) | n (%) | n (%) | n (%) |
| Posterior Subcapsular | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) | n (%) | n (%) |
| Grade | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| +1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| +2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| +3 | n (%) | n (%) | n (%) | n (%) | n (%) |
| +4 | n (%) | n (%) | n (%) | n (%) | n (%) |
| hath Caharta 1 and 2 | ` ' | | ` ' | * * | • / |

path\t program.sas date

Programmer Note: Continue table for Eyelashes, Conjunctiva, Sclera, Cornea, Anterior Chamber Flare), Iris, Lens Status, Cataract Type, Grade..

Programmer Note: Continue table for Visits: Day1, Day2, Day3, Day7, Day14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term.

Total includes both Cohorts 1 and 2.

[2] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

<sup>[3]</sup> Subject may be counted more than one row.

Programmer Note: Table 14.3.4.6.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

Programmer Note: Table can be modified to align with information collected on the CRF.

jCyte, Inc. Page 1 of x Protocol: JC-01

**Table 14.3.4.7** Fundus Photography by Eye Vitreous Examination **Safety Population** 

| | Cohort 1 | | Cohort | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Study Eye | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| | | ••• | | ••• | |
| Non-Study Eye | | | | | |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

Table 14.3.4.8.1 Intraocular Pressure (IOP): Study Eye Safety Population

| | Coho | ort 1 | Coho | Cohort 2 | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | •••• | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | (N=) | | | (N=) |
| Baseline [2] | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1 | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) |
| Median | xx.x | XX.X | XX.X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 1 Change from Baseline | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 2 | | | | | |
| n | n | n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x(xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx |
| •• | | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Day 3, Day 7, Day14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term. Programmer Note: Table 14.3.4.8.2 will contain the same information for the Non-Study Eye.

Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

**Table 14.3.4.9.1 B-Scan: Study Eye Safety Population** 

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Good | n (%) | n (%) | n (%) | n (%) | n (%) |
| Poor | n (%) | n (%) | n (%) | n (%) | n (%) |
| Injected Cells Visualized | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 3 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Good | n (%) | n (%) | n (%) | n (%) | n (%) |
| Poor | n (%) | n (%) | n (%) | n (%) | n (%) |
| Injected Cells Visualized | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) | n (%) | n (%) |
| both Cohorts 1 and 2 | | | | | |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

path\t\_program.sas date

Programmer Note: Continue table for Visits: Day 7, Month3, Month 6, Month 12/Early Term.

Programmer Note: Table 14.3.4.9.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit.

Table 14.3.4.10.1 Dilated Fundoscopic Examination: Study Eye **Safety Population** 

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | •••• | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Vitreous Examination | | | . , | | . , |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Very Severe +4 | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Very Severe +4 | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Day 2 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) | n (%) | n (%) |
| Very Severe +4 | | | | | |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Optic Nerve, Macula, and Peripheral Retina Examinations.

Programmer Note: Continue table for Visits: Day 3, Day 7, Day 14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term.

Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

Programmer Note: Table 14.3.4.10.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

**Table 14.3.4.11** Post Injection Clinical Vitreous Exam: Study Eye **Safety Population** 

| | Cohort | : 1 | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Day0 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Injected eye examined | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Methods of Examination [2] | | | | | |
| Indirect Ophthalmoscopy | n (%) | n (%) | n (%) | n (%) | n (%) |
| Fundus Exam | n (%) | n (%) | n (%) | n (%) | n (%) |
| Slit Lamp Exam | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) |
| Change from Previous Exam | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Appearance | | | | | |
| Cells | n (%) | n (%) | n (%) | n (%) | n (%) |
| Clumps | n (%) | n (%) | n (%) | n (%) | n (%) |
| Opacity | n (%) | n (%) | n (%) | n (%) | n (%) |
| Debris | n (%) | n (%) | n (%) | n (%) | n (%) |
| Strands | n (%) | n (%) | n (%) | n (%) | n (%) |
| Inflammation | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) |
| Photograph taken | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |

path\t program.sas date

Programmer Note: Continue table for Visits: Day 1, Day 2, Day 3, Day 7, Day 14, Day 21, Day 28, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12/Early Term. Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] Subject may be counted more than one row.

Table 14.3.4.12.1 Optical Coherence Tomography (OCT): Study Eye **Categorical Analysis** ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | •••• | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup><br>(N=) |
| Cystoid Macular Edema (CME) present | | | | | |
| Baseline [2] | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Day 28 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 3 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 9 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 12/ Early Termination | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| If CME Present, Involve Foveal Center | | | | | |
| Baseline [2] | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Day 28 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 3 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 9 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 12/ Early Termination | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Month 6, Month 9, Month 12/Early Term.

Programmer Note: Table 14.3.4.12.2 will contain the same information for the Non-Study Eye.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date time

## Table 14.3.4.13.1 Fluorescein Angiography: Study Eye Categorical Analysis ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | 0.5 x 10 <sup>6</sup> hRPC<br>(N=) | | Total <sup>[1]</sup> (N=) |
| Active Leakage | | | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 12/ Early Termination | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Ischemia | | | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| Month 12/ Early Termination | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |

<sup>[1]</sup> Total includes both Cohorts 1 and 2.

Programmer Note: Continue table for Visits: Month 6, Month 9, Month 12/Early Term.

Programmer Note: for Active Leakage and Ischemia present for "YES"

Programmer Note: Table 14.3.13.2 will contain the same information for the Non-Study Eye.

<sup>[2]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Table 14.3.4.14.1 **Autofluorescence: Study Eye** ITT Population

| | Cohort 1 | | Cohort 2 | | |
|---|---|---|---|---|---|
| | 0.5 x 10 <sup>6</sup> hRPC | | 0.5 x 10 <sup>6</sup> hRPC | | Total [1] |
| | (N=) | | (N=) | | (N=) |
| Baseline [2] | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Month 12/ Early Termination | (n=) | (n=) | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) | n (%) | n (%) |

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point. Programmer Note: Table 14.3.4.14.2 will contain the same information for the Non-Study Eye.

<sup>[1]</sup> Total includes both Cohorts 1 and 2.
[2] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

Appendix D: Listing Layouts

Page 1 of x jCyte, Inc. Protocol: JC-01

## Listing 16.2.1.1 Subject Disposition

| Treatment Group | Subject<br>ID | Safety<br>Population <sup>[1]</sup> | ITT Population [2] | Information Consent<br>Date | First Drug<br>Administration<br>Date/Time | Completion or Discontinuation Date | Primary Reason for Discontinuation |
|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | Yes/No | Date9. | Date9./time5. | Date9. | xxxxxxxxxxxxxx |
| | <br>xxxxxx | <br>Yes/No<br> | Yes/No | Date9. | Date9./time5. | Date9. | xxxxxxxxxxxxxx |

Programmer Note: Include Reasons, Death and AE # information in "Primary Reason for Discontinuation" column.

<sup>[1]</sup> Received any amount of jCell treatment.
[2] All enrolled subjects who provide any post-screening data.
path\l\_program.sas date time

jCyte, Inc.
Protocol: JC-01

## Listing 16.2.2.1 Protocol Deviations

| Treatment Group | Subject<br>ID | Deviation Type | Protocol Deviation Category | Description of Protocol Deviation |
|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | XXXXXX | xxxxxxxx | xxxxxxxx |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | xxxxxx | xxxxxxxx | xxxxxxxx |

path\l\_program.sas date time
jCyte, Inc. Protocol: JC-01

### Listing 16.2.2.2 Inclusion/Exclusion Criteria

| Treatment Group | Subject<br>ID | All Eligibility<br>Criteria Met? | If Not Met,<br>Inc/Exc Criterion ID Not Met | Protocol Version Date |
|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Yes/No | Inclusion #/Exclusion# | Date9. |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | Inclusion #/Exclusion# | Date9. |

path\l\_program.sas date time

Protocol: JC-01

# Listing 16.2.4.1 Demographic and Baseline Characteristics

| Treatment Group | Subject ID | Date of<br>Birth | Age<br>(years) | Sex | If Female,<br>Childbearing<br>Potential? | If YES,<br>Method of<br>Birth Control | Ethnicity | Race | Previously Typed to Determine PR Gene Mutation? | Study<br>Eye | Baseline<br>Height<br>(cm) | Baseline<br>Weight<br>(Kg) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Date9. | xx | Female | No/Yes | IUD | Hispanic or Latino | White | Yes/No | OD(Right) | xxx | xxx |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Date9. | XX | Male | No/Yes | Oral<br>Contraception | Not<br>Hispanic<br>or Latino | Asian | Yes/No | OS(Left) | XXX | xxx |
| ••••• | | | | | | | | | | | | |

path\l\_program.sas date time

Programmer Note: Include Specification for Other in "Method of Birth Control" column if applicable

#### **Listing 16.2.4.2 Medical History**

| Treatment Group | Subject ID | Past Diseases or Surgeries? | MH# | Body System | Medical History Condition/Event | Start Date | End Date/Ongoing |
|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | 1 | xxxxxxx | xxxxxxxxxx | Date9. | Date9./Ongoing |
| | ••••• | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | 2 | xxxxxxx | xxxxxxxxxxx | Date9. | Date9./Ongoing |

path\l program.sas date time

Programmer Note: sort by medical history number within each subject.
Programmer Note: If MH marked as Ongoing, then show "Ongoing" under End Date column.

jCyte, Inc. Protocol: JC-01

#### **Listing 16.2.4.3** Ocular Medical History

| Treatment Group | Subject ID | Ocular Medical<br>History? | Ocular<br>MH # | Eye | Body System | Ocular MH<br>Condition/Diagnosis/Surgery | Date of<br>Diagnosis/Surgery | Date Resolved/Ongoing |
|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Yes/No | 1 | OD | xxxxxxxxxxx | xxxxxxxxxxx | Date9. | Date9./Ongoing |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | 1 | OS | xxxxxxxxxxx | xxxxxxxxxxx | Date9. | Date9./Ongoing |

path\l\_program.sas date time

Programmer Note: sort by medical history number within each subject.

Programmer Note: If MH marked as Unknown start or end date, then show "Unknown" under Date of Diagnosis/Surgery or Date Resolved columns, respectively. Programmer Note: If MH marked as Ongoing end date, then show "Ongoing" under Date Resolved column.

### Listing 16.2.4.4 Urine Drug Screen

| Treatment Group | Subject ID | Visit | Collection Date | Collection<br>Time | Any Test<br>Results Positive? | If YES, Which Tests<br>Were Positive? |
|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening | Date9. | Time5. | Yes/No | Test Name |
| Cohort 1 – 1.0 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening | Date9. | Time5. | Yes/No | Test Name |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening | Date9. | Time5. | Yes/No | Test Name |
| Cohort 2 – 1.0 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening | Date9. | Time5. | Yes/No | Test Name |

.....

path\l\_program.sas date time

### Listing 16.2.4.5 Infectious Disease Tests

| Treatment Group | Subject ID | Visit | Tested for<br>Hepatitis B:<br>Reason | Hepatitis B<br>Result | Tested for<br>Hepatitis C?<br>Reason | Hepatitis C<br>Result | Tested for HIV? Reason | HIV<br>Result |
|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening<br>Baseline | Yes<br>No: Reason | Negative/Positive | Yes<br>No: Reason | Negative/Positive | Yes<br>No: Reason | Negative/Positive |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening<br>Baseline | Yes<br>No: Reason | Negative/Positive | Yes<br>No: Reason | Negative/Positive | Yes<br>No: Reason | Negative/Positive |

path\l\_program.sas date time

.

Listing 16.2.5.1 Study Drug Administration

| | | | | | | | | | | | IOP | Prescribed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | AEs | Vital Signs | Measurement | Topical |
| | | | | | | | | | Observed? | comparable to | less than 30 mm | Treatment af |
| | | | | | | Eye Drug | Total Dose | Dose | | Pre-Treatment of | f Post Treatment | Treatment o |
| Treatment | Subject ID | | Administration | Dilation | Injection | | | l Interruptions? | | Study drug | of Study Drug | Study Drug |
| Group | (Study Eye) | Visit | Date | Time | Time | Into | ? Reason | Reason | | Injection | Injection | Injection |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | Xxxxx (OS) | Day 0 | Date 9. | Time5. | Time5. | OS (Left) | Yes | Yes: Reason | No/Yes | No/Yes | No/Yes | No/Yes |
| Cohort 1 - 1.0 x<br>10 <sup>6</sup> hRPC | Xxxxx (OD) | Day 0 | Date9. | Time5. | Time5. | OD<br>(Right) | No: Reason | No | No | No | No | No |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | Xxxxx (OS) | Day 0 | Date9. | Time5. | Time5. | OS (Left) | Yes | Yes: Reason | No/Yes | No/Yes | No/Yes | No/Yes |
| Cohort 2 - 1.0 x<br>10 <sup>6</sup> hRPC | Xxxxx (OD) | Day 0 | Date9. | Time5. | Time5. | OD<br>(Right) | No: Reason | No | No | No | No | No |

Listing 16.2.6.1
Best Corrected Visual Acuity (ETDRS)

| | | | Assessment | OD Visual | Acuity | OS Visual Acuity | |
|---|---|---|---|---|---|---|---|
| Treatment Group | Subject<br>ID | Visit | Assessment Date (Study Day) | Measurement | Total Numbers of<br>Letters Missed | Measurement | Total Numbers of<br>Letters Missed |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | Screening | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Baseline | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day0 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day1 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day2 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day3 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day7 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day14 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day21 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Day28 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month2 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month3 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month4 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month6 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month9 | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | XXX |
| | | Month12 or<br>Early<br>Termination | Date9. (xx) | Xx/xxx | xxx | Xx/xxx | XXX |
| Cohort 1 - 1.0 x 10 <sup>6</sup> hRPC | xxx-xxx | | Not Done:<br>Reason | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxx-xxx | | Date9. (xx) | Xx/xxx | XXX | Xx/xxx | xxx |
| Cohort 2 - 1.0 x 10 <sup>6</sup> hRPC | xxx-xxx | | Date9. (xx) | Xx/xxx | xxx | Xx/xxx | xxx |
| date time | | | | | | | |

path\l\_program.sas date tii

Programmer Note: If NO marked for testing, include reason in "Assessment Date" column.

#### Listing 16.2.6.2.1 Electroretinogram Right Eye (OD)

Dark Adapted 0.01 ERG (Rod Response)

| | | | | | | | Dark | Adapted 0.01 | LICO (ICOU ICESPO | J118C) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ERG Prior to | ERG | | | | | Time from | Time from | | If Abnormal, | |
| | | | Ancillary | Date (Study | Start | Stop | A-Wave | B-Wave | Flash to A- | Flash to B- | | Change from | |
| Treatment Group | Subject ID | Visit | Testing? | Day) | Time | Time | Amplitude | Amplitude | Wave Trough | Wave Peak | Result | Previous Visit | Abnormality |
| Cohort 1 - 0.5 x 10 <sup>6</sup><br>hRPC | XXXXXX | Screening | Yes/No | Date9. (xx) | Time5. | Time5. | | | | | Normal | | |
| | | Baseline | Yes/No | Date9. (xx) | Time5. | Time5. | | | | | Abnormal CS | Yes/No | XXXXXXXX |
| | | Month6 | Yes/No | Not Done: | Time5. | Time5. | | | | | Abnormal NCS | Yes/No | XXXXXXXX |
| | | | | reason | | | | | | | | | |
| | | Month12 | | | | | | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup><br>hRPC | xxxxxx | Screening | Yes/No | Date9. (xx) | Time5. | Time5. | | | | | Normal | | |
| | | Baseline | Yes/No | Date9. (xx) | Time5. | Time5. | | | | | Abnormal NCS | Yes/No | XXXXXXXX |
| | | Month6<br>Month12 | Yes/No | Date9. (xx) | Time5. | Time5. | | | | | Abnormal CS | Yes/No | xxxxxxxx |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

. . . . . .

path\l program.sas date time

Programmer Note: If NO marked for testing, include reason in "ERG Date" column.

Programmer Note: Include Description of Abnormality and Clinically Significant information in "Result" column.

Programmer Note: Repeat columns for Dark Adapted 3.0 ERG (Rod Cone Response), Light Adapted 3.0 (Single Rod Cone Response), Light Adapted 3.0 Flicker ERG.

Programmer Note: 16.2.6.2.2 Repeat same for left Eye columns for Dark Adopted 0.01 ERG (rod response), Dark Adapted 3.0 ERG (Rod Cone Response), Light Adapted 3.0 (Single Rod Cone Response),

Light Adapted 3.0 Flicker ERG.

Listing 16.2.6.3 Optical Coherence Tomography (OCT)

| Treatment Group | Subject ID | Visit | Assessment<br>Date (Study<br>Day) | Cystoid Macular Edema<br>(CME) Present? | IF CME Present, Involve<br>Foveal Center? | OD Central Subfield<br>Thickness (um) | OS Central Subfield<br>Thickness (um) |
|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline Day 28 Month 3 Month 6 Month 12 or Early Termination | Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) | Yes/No<br>Yes/No<br>Yes/No<br>Yes/No<br>Yes/No | Yes/No<br>Yes/No<br>Yes/No<br>Yes/No | XXX<br>XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX<br>XXX |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx<br> | Baseline Day 28 Month 3 Month 6 Month 12 or Early Termination | Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) | Yes/No<br>Yes/No<br>Yes/No<br>Yes/No<br>Yes/No | Yes/No<br>Yes/No<br>Yes/No<br>Yes/No<br>Yes/No | XXX<br>XXX<br>XXX<br>XXX<br>XXX | XXX<br>XXX<br>XXX<br>XXX<br>XXX |

path\l\_program.sas date time

Programmer Note: If NO marked for testing, include reason in "Assessment Date" column.

Protocol: JC-01

# Listing 16.2.6.4 Fluorescein Angiography

| | | | | | | OD | (Right) | | | OS (Left) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Assessment | | | Active | | Other | | Active | | Other |
| Treatment Group | Subject ID | Visit | Date(Study Day) | Imaging Type | Start Time | Leakage? | Ischemia? | Observations | Start Time | Leakage? | Ischemia? | Observations |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | Date9. (xx) | Field Imaging | Time5. | Yes/No | Yes/No | XXXXXX | Time5. | Yes/No | Yes/No | xxxxxx |
| | | Month 6 | Date9. (xx) | Wide Field Imaging | Time5. | Yes/No | Yes/No | XXXXXX | Time5. | Yes/No | Yes/No | XXXXXX |
| | | Month 12 | Date9. (xx) | Other: specify | Time5. | Yes/No | Yes/No | XXXXXXX | Time5. | Yes/No | Yes/No | XXXXXXX |
| Cohort 2 - 0.5 x 10 <sup>6</sup><br>hRPC | XXX | Baseline | Date9. (xx) | Field Imaging | Time5. | Yes/No | Yes/No | XXXXXXX | Time5. | Yes/No | Yes/No | XXXXXXX |
| | | Month 6<br>Month 12 | | Wide Field Imaging<br>Other | Time5.<br>Time5. | Yes/No<br>Yes/No | Yes/No<br>Yes/No | XXXXXXX<br>XXXXXX | Time5.<br>Time5. | Yes/No<br>Yes/No | Yes/No<br>Yes/No | XXXXXXX<br>XXXXXX |

. . . . . .

path\l\_program.sas date time

Programmer Note: If NO marked for testing, include reason in "Assessment Date" column.

#### Listing 16.2.6.5 Autofluorescence

| | | | | | | Abnormal, | | Abnormal, |
|---|---|---|---|---|---|---|---|---|
| | | | | Pupils Dilated | | Change from | | Change from |
| | | | Assessment | for Imagining | Right Eye | Previous Visit? | Left Eye (OS) | Previous Visit? |
| Treatment Group | Subject ID | Visit | Date (Study Day) | Exam? | (OD) Result | | Result | |
| 6 | | | | | | | | |
| Cohort 1 - $0.5 \times 10^6 \text{ hRPC}$ | XXXXXX | Baseline | Date9. (xx) | Yes/No | Normal | | Normal | |
| | | Month 6 | Not Done: reason | Yes/No | Abnormal CS: | Yes | Abnormal | Yes |
| | | | | | Abnormality | | CS:Abnoramlity | |
| | | Month 12 or Early | Date 9. (xx) | Yes/No | Abnormal | No | Abnormal NCS | No |
| | | Termination | | | NCS: | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Baseline | Date9. (xx) | Yes/No | Normal | | Normal | |
| Conort 2 - 0.5 x 10 mg C | AAAAAA | Month 6 | Date9. (xx) | Yes/No | | Not Applicable | | Not Applicable |
| | | Wolldi O | Dates. (XX) | 1 65/110 | Abnormality | Not Applicable | Abnormality | Not Applicable |
| | | Month 12 or Early | Date9. (xx) | Yes/No | Abnormal | No | Abnormal NCS | No |
| | | Termination | | | NCS | | | |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time

Programmer Note: If NO marked for testing, include reason in "Assessment Date" column.

Programmer Note: Include Description of Abnormality and Clinically Significant information in "Result" column

### Listing 16.2.6.6 Visual Field Examination

| | | | | | | | | | OD (Rig | ght) | | | | O: | S (Left) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Pupil<br>Dialated<br>Assessment | | Overall Comments | i | If<br>Abnormal,<br>Change | | | | | | If Abnormal, Change from Baseline | | | | False | e |
| Treatment<br>Group | Subject<br>ID | Visit | Date (study<br>Day) | Visual Field<br>Technology | | Result | from<br>Baseline | Mean<br>Dev. | Fixation<br>Loss | False<br>Positive | False<br>Negative | Result | | Mean<br>Dev. | | n False<br>Positive | | iv<br>— |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | Date9. (xx) Yes | Goldmann<br>VF | xxxxxxxx | Normal | | | | | | Normal | | | | | | |
| ma c | | Month 6 | Date9. (xx) | Humphrey<br>10-2 | XXXXXXXX | Abnormal<br>NCS | Yes | | | | | Abnormal<br>NCS | No | | | | | |
| | | Month 12 of<br>Early<br>Termination | orNot Done:<br>Reason<br>n | 10 2 | | THES | | | | | | Nes | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | Date9. (xx) No | Other: | xxxxxxxx | Normal | | | | | | Normal | | | | | | |
| ind C | | Month 6 | Date9. (xx) | Goldmann<br>VF | xxxxxxxx | Normal | | | | | | Normal | | | | | | |
| | | Month 12 c<br>Early<br>Termination | orDate9. (xx) | Humphrey<br>10-2 | xxxxxxxx | Normal | | | | | | Abnormal<br>Cs | Not<br>Applicable | | | | | |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time

Programmer Note: If NO marked for testing, include reason in "Assessment Date" column.

Programmer Note: Include Description of Abnormality and Clinically Significant information in "Result" column

Listing 16.2.7.1 Adverse Events

| | | Verbatim Term | // | Onset Time | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | System Organ | | | | | | Relationship | | |
| Treatment | Subject | Class//Preferred | Onset Date | | End Date | | | to Study | Treatment | |
| Group | ID | AE# Term | (Study Day) | | (Study Day) | Serious | Severity | Drug | of Event | Outcome |
| Cohort 1 - 0.5 x | XXXXXX | | Date9.(xx) | Time5. | Date9.(xx) | Yes | Mild | Not Related | None | Recovery/Resolved |
| 10 <sup>6</sup> hRPC | | | | | | | | | | |
| | | | Date9.(xx) | Time5. | Date9.(xx) | No | Moderate | Unlikely | Medication | Recovery/Resolved W/Seq |
| | | | | | | | | Related | | |
| | | | Date9.(xx) | Time5. | Date9.(xx) | No | Moderate | Possibly | Non-Drug | Recovering/Resolving |
| | | | | | | | | Related | Treatment | |
| | | | Date9.(xx) | | Date9.(xx) | No | Mild | Related | Hospitalization | |
| | | | Date9.(xx) | | Date9.(xx) | No | Severe | Unlikely | | |
| | | | | | | | | Related | | |
| | | | Date9.(xx) | | Date9.(xx) | No | Mild | | | |

Cohort 2 - 0.5 x xxx--xxx 10<sup>6</sup> hRPC

path\l\_program.sas date time

Programmer Note: sort by subject and AE # subject

jCyte, Inc. Protocol: JC-01

# Listing 16.2.7.2 Serious Adverse Events

Verbatim Term //

| Treatment Group | Subject<br>ID | System Organ AE Class//Preferred # Term | Onset Date<br>(Study Day) | Onset<br>Time | End Date<br>(Study Day) | Severity | Relationship<br>to Study Drug | Treatment of Event | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | 110 | ,, 101111 | (Study Buy) | Time | (Study Buy) | Sevening | to Study Drug | or Event | Guicome |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | | Date9.(xx) | Time5. | Date9.(xx) | Mild | Not Related | None | Recovery/Resolve d |
| | | | Date9.(xx) | | Date9.(xx) | Moderate | Unlikely<br>Related | Medication | Recovery/Resolve<br>d W/Seq |
| | | | Date9.(xx) | | Date9.(xx) | Moderate | Possibly<br>Related | Non-Drug<br>Treatment | Recovering/Resol ving |
| | | | Date9.(xx) | | Date9.(xx) | Mild | Related | Hospitalization | |
| | | | Date9.(xx) | | Date9.(xx) | Severe | Unlikely<br>Related | • | |
| | | | Date9.(xx) | | Date9.(xx) | Mild | | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

.....

.....

path\l\_program.sas date time

Programmer Note: sort by subject and AE # subject

#### **Listing 16.2.7.3** Related Adverse Events

| | Subject | ΑE | | Onset<br>Date/Time | End Date | | | Relationship | Treatment | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | ID | # | Verbatim Term // Preferred Term | (Study Day) | (Study Day) | Serious | Severity | to Study Drug | of Event | Outcome |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | | | Date9.(xx) | Date9.(xx) | Yes | Mild | Related | None | Recovery/Resolved |
| | | | | Date9.(xx) | Date9.(xx) | No | Moderate | Related | Medication | Recovery/Resolved<br>W/Seq |
| | | | | Date9.(xx) | Date9.(xx) | No | Moderate | Possibly Related | Non-Drug<br>Treatment | Recovering/Resolving |
| | | | | Date9.(xx) | Date9.(xx) | No | Mild | Related | Hospitalizat ion | |
| | | | | Date9.(xx)<br>Date9.(xx) | Date9.(xx)<br>Date9.(xx) | Yes<br>No | Severe<br>Mild | Related | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

.....

path\l\_program.sas date time

.....

Programmer Note: sort by subject and AE # subject Programmer Note: include Onset Time if available in Onset Date column.

Listing 16.2.7.4 Post Injection Clinical Vitreous Exam

| Treatment Group | Subject ID | Visit | Examination<br>Date (Study<br>Day) | Method<br>Used | Change<br>from Prev.<br>Visit | Appearance | Size | Location | Photograph<br>Taken? |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Day 0 | Date9.(xx) | Indirect | Yes/No | Cells | xxxxxx | xxxxxx | Yes/No |
| | | D 1 | D ( 0 ( ) | Ophthalmoscopy | 37 /NT | CI | | | 37 /3T |
| | | Day 1 | Date9.(xx) | Fundus Exam | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Day 2 | Date9.(xx) | Slit Lamp Exam | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | Day 3 | Date9.(xx) | Other: | Yes/No | Debris | XXXXXX | XXXXXX | Yes/No |
| | | Day 7 | Date9.(xx) | Indirect<br>Ophthalmoscopy | Yes/No | Stands | XXXXXX | XXXXXX | Yes/No |
| | | Day 14<br>Day 21 | Date9.(xx)<br>Not Done: | Fundus Exam | Yes/No | Inflammation | XXXXXX | XXXXXX | Yes/No |
| | | | Reason | | | | | | |
| | | Day 28 | Date9.(xx) | Other: | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Month 2 | Date9.(xx) | Indirect<br>Ophthalmoscopy | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | Month 3 | Date9.(xx) | Fundus Exam | Yes/No | Debris | XXXXXX | XXXXXX | Yes/No |
| | | Month 4 | Date9.(xx) | Slit Lamp Exam | Yes/No | Stands | XXXXXX | XXXXXX | Yes/No |
| | | Month 5 | Date9.(xx) | Other: | Yes/No | Inflammation | XXXXXX | XXXXXX | Yes/No |
| | | Month 9 | Date9.(xx) | Slit Lamp Exam | Yes/No | Cells | XXXXXX | XXXXXX | Yes/No |
| | | Month 12 or<br>Early<br>Termination | Date9.(xx) | Other: | Yes/No | Other: | XXXXXX | XXXXXX | Yes/No |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | | | | | | | | |

path\l\_program.sas date time

Programmer Note: If NO marked for examination, include reason in "Examination Date" column. Methods used include all applicable Methods.

#### Listing 16.2.8.1 Hematology Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date (Study<br>Day) | Collection Time | Hemoglobin<br>(g/dL) | Hematocrit (%) | Platelet Count (x 10^3/uL) | Red Cell Count<br>(x 10^6/uL) | White Cell Count (x 10^3/uL) |
|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup><br>hRPC | XXXXX | x Screening | Date9. (xx) | Time5. | | | | | |
| | | Baseline | Date9. (xx) | Time5. | | | | | |
| | | Day 7 | Date9. (xx) | Time5. | | | | | |
| | | Day 28 | Date9. (xx) | Time5. | | | | | |
| | | Month 3 | Date9. (xx) | Time5. | | | | | |
| | | Month 6 | Date9. (xx) | Time5. | | | | | |
| | | Month 12 or | Date9. (xx) | Time5. | | | | | |
| | | Early | ` ′ | | | | | | |
| | | Termination | | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> | XXXXX | x | | | | | | | |

Listing 16.2.8.1 Hematology Part 2 of 2

Lymphocytes Lymphocytes Eosiophils Subject Neutrophils (%) Monocytes Eosinophils Basophils Neutrophils (x 10^3/uL) Monocytes Basophils Collection  $(x 10^3/uL)$ Treatment Group ID Visit Date/Time (%)(%)(%) (%)  $(x 10^3/uL)$  $(x 10^3/uL)$  $(x 10^3/uL)$ 

Note: L=Low and H=High, CS=Clinically Significant

hRPC

Programmer Note: If NO marked for examination, include reason in "Examination Date" column.

. path\l\_program.sas date time

**Listing 16.2.8.2** Chemistry Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date (Study<br>Day) | Collection<br>Time | Sodium<br>(mmol/L)) | Potassium<br>(mmol/L) | Chloride<br>(mmol/L) | Bicarbonate (mmol/L) | ALT<br>(U/L) | AST<br>(U/L) | Alkaline<br>Phosphatase<br>(U/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Screening Baseline Day 7 Day 28 Month 3 Month 6 Month 12 or Early Termination | Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) Not Done: Reason Date9. (xx) Date9. (xx) | Time5. Time5. Time5. Time5. Time5. | | | | | | | |

Cohort 2 - 0.5 x 10<sup>6</sup> hRPC xxx--xxx

Listing 16.2.8.2 Chemistry Part 2 of 2

| | | | Collection | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject | | Date (Study | Collection | BUN | Creatinine | Total Protein | Albumin | Calcium | Phosphate | Glucose |
| Treatment Group | ID | Visit | Day) | Time | (mg/dL) | (mg/dL) | (g/dL) | (g/dL) | (mg/dL) | (mg/dL) | (mg/dL) |

Cohort 1 - 0.5 x 10<sup>6</sup> hRPC xxx--xxx Screening Date9. (xx) Time5.

Note: L=Low and H=High, CS=Clinically Significant.

path\l\_program.sas date

time

#### Listing 16.2.8.3 Coagulation

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date/ (Study<br>Day) | Collection<br>Time | PT (sec) | PTT (sec) | INR | Coagulation Results Abnormal?/if Yes:<br>Abnormatlity |
|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | | Canaanina | Data() (vv) | Time5 | | | | Yes: NCS |
| Conort 1 - 0.3 x 10° nRPC | XXXXXX | Screening<br>Baseline | Date9. (xx)<br>Date9. (xx) | Time5.<br>Time5. | | | | Yes: NCS |
| | | Day 7 | Date 9. (xx) | Time5. | | | | No |
| | | Day 7<br>Day 28 | Date9. (xx) | Time5. | | | | Yes: CS |
| | | 2 | ( ) | | | | | ies. Cs |
| | | Month 3 | Date9. (xx) | Time5. | | | | |
| | | Month 6 | Date9. (xx) | Time5. | | | | |
| | | Month 12 or | Date9. (xx) | Time5. | | | | |
| | | Early | | | | | | |
| | | Termination | | | | | | |
| | •••• | | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | | | | | | | |

.....

Note: CS=Clinically Significant. path\l\_program.sas date time

Programmer Note: Include Clinically Significant information in "Coagulation Results Abnormal?" column.

#### Listing 16.2.8.4 Urinalysis Part 1 of 2

| | Subject | | Collection Date (Study | Collection | Specific | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | ID | Visit | Day) | Time | Gravity | рН | Glucose | Bilirubin | Ketone | Blood | Protein | Urobilinogen |
| Cohort 1 - 0.5 x 10 <sup>6</sup><br>hRPC | xxxxxx | Screening | Date9. (xx) | Time5. | | | Negative | Negative | Negative | Negative | Negative | Negative |
| | | Baseline | Date9. (xx) | Time5. | | | positive | positive | positive | positive | positive | positive |
| | | Month 3 | Date9. (xx) | Time5. | | | Negative | Negative | Negative | Negative | Negative | Negative |
| | | Month 6 | Not Done,<br>Reason: | | | | S | 2 | 2 | 2 | Ü | S |
| | | Month 12 or<br>Early | Date9. (xx) | Time5. | | | positive | positive | positive | positive | positive | positive |
| | | Termination | | | | | | | | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup><br>hRPC | xxxxxx | | | | | | | | | | | |

#### Listing 16.2.8.4 Microscopic Exam Part 2 of 2

| | | | | | Mic | croscopic Exam | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Visit | Collection Date (Study Day) | Collection Time | WBC<br>(/hpf) | RBC<br>(/hpf) | Enithelial Cells | Bacteria | Other |
| xxxxx | Screening | Date9. (xx) | Time5. | | | 1 | Absent/Present | |
| | IĎ | ID Visit | ubject Date (Study ID Visit Day) | abject Date (Study ID Visit Day) Collection Time | ubject Date (Study WBC ID Visit Day) Collection Time (/hpf) | Collection Libject Date (Study WBC RBC LD Visit Day) Collection Time (/hpf) (/hpf) | Collection ubject Date (Study WBC RBC ID Visit Day) Collection Time (/hpf) (/hpf) Epithelial Cells | Collection ubject Date (Study WBC RBC ID Visit Day) Collection Time (/hpf) (/hpf) Epithelial Cells Bacteria |

path\l\_program.sas date time

jCyte, Inc. Protocol: JC-01

## **Listing 16.2.8.5** Clinically Significant Lab Values Part 1 of 2

| Treatment Group | Subject ID | Visit | Collection<br>Date (Study Day) | Collection Time | Lab Category | Lab Test | Value |
|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup><br>hRPC | xxxxxx | Screening | Date9. (xx) | Time5. | Hematology | Hemoglobin | |
| | | Baseline | Date9. (xx) | Time5. | | Hematocrit | |
| | | Month 3 | Date9. (xx) | Time5. | | | |
| | | Month 6 | Not Done, Reason: | | | | |
| | | Month 12 or Early<br>Termination | Date9. (xx) | Time5. | | | |
| Cohort 2 - 0.5 x 10 <sup>6</sup><br>hRPC | xxxxxx | | | | Chemistry | Albumin | |

path\l\_program.sas date time

Programmer Note: Include only Clinically Significant Abnormal values from all Lab tests.

Listing 16.2.8.6 Vital Signs

| <b>T</b> | G 1. | | Measurement | | | CDD/DDD | | Respiration | <b>.</b> | **** | TT 1.1. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | *** | Date (Study | | | SBP/DBP | Heart Rate | Rate | Temperature | Weight | Height |
| Group | ID | Visit | Day) | Time | Time Point | (mmHg) | (beats/min) | (breaths/min) | (C) | (Kg) | (cm) |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening | Date9.(xx | Time5. | | Xxx/xxx | xxx | xxx | XXX | xxx | XXX |
| | | Baseline | Date9.(xx | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | Date9.(xx) | Time5. | 15 min Pre-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | J | Date9.(xx) | Time5. | 15 min Post-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | | Date9.(xx) | Time5. | 60 min Post-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 1 | Date9.(xx) | Time5. | v | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 2 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 3 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 7 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 14 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 21 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 28 | Not Done:<br>Reason | | | | | | | | |
| | | Month 2 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 3 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 4 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 5 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 9 | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 12 or | Date9.(xx) | Time5. | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Early | . , | | | | | | | | |
| | | Termination | | | | | | | | | |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Day 0 | Date9.(xx) | Time5. | | | | | | | |

path\l\_program.sas date time

Listing 16.2.8.7.1 12-Lead Electrocardiogram

| Treatment Group | Subject<br>ID | Visit | ECG Date<br>(Study Day) | ECG<br>Time | Subject<br>Position | Interpretation | Heart Rate (bpm) | RR<br>(msec) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcB<br>(msec) | QTcF<br>(msec) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | Screening | Date9.(xx | Time5. | Sitting | Normal | XX | xxxx | XXX | XX | XXX | XX.XX | xxx.xx |
| | | Baseline | Date9.(xx | Time5. | Standing | Abnormal CS | XX | XXXX | XXX | XX | XXX | xx.xx | XXX.XX |
| | | Day 0 | Date9.(xx) | Time5. | Supine | Normal | XX | XXXX | XXX | XX | XXX | XX.XX | XXX.XX |
| | | Day 1 | Date9.(xx) | Time5. | Prone | Abnormal | XX | XXXX | XXX | XX | XXX | XX.XX | XXX.XX |
| Cohort 2 - $0.5 \text{ x}$<br>$10^6 \text{ hRPC}$ | XXXXXX | Screening | Date9.(xx | Time5. | Sitting | Normal | XX | xxxx | XXX | XX | XXX | XX.XX | XXX.XX |
| | | Baseline | Date9.(xx | Time5. | Standing | Abnormal NCS | XX | XXXX | XXX | XX | XXX | XX.XX | XXX.XX |
| | | Day 0 | Date9.(xx) | Time5. | Supine | Normal | XX | XXXX | XXX | XX | XXX | XX.XX | XXX.XX |
| | | Day 1 | Date9.(xx) | Time5. | Prone | Abnormal NCS | XX | XXXX | XXX | XX | XXX | XX.XX | XXX.XX |

.....

Note: CS=Clinically Significant, NCS=Not Clinically Significant. path\l\_program.sas date time

Programmer Note: If NO marked for ECG, include reason in "ECG Date/Time" column.

Listing 16.2.8.7.2 Clinically Significant 12-Lead Electrocardiogram Interpretation

| Treatment Group | Subject<br>ID | Visit | ECG Date<br>(Study Day) | ECG Time | Subject<br>Position | Interpretation |
|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening<br>Baseline<br>Day 1 | Date9.(xx<br>Date9.(xx<br>Date9.(xx) | Time5. Time5. Time5. | Sitting<br>Standing<br>Prone | AbNormal CS<br>Abnormal CS<br>Abnormal CS |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening<br>Baseline<br>Day 0<br>Day 1 | Date9.(xx<br>Date9.(xx<br>Date9.(xx)<br>Date9.(xx) | Time5. Time5. Time5. Time5. | Sitting<br>Standing<br>Supine<br>Prone | AbNormal CS<br>Abnormal CS<br>AbNormal CS<br>Abnormal CS |

.....

Note: CS=Clinically Significant. path\l\_program.sas date time

Programmer Note: If NO marked for ECG, include reason in "ECG Date/Time" column.

#### Listing 16.2.8.8 Physical Examination

| Treatment Group | Subject<br>ID | Visit | Examination Date (Study Day) | Were There Any<br>Abnormal Findings on<br>the Physical Exam? | Any Changes in Vision or Light<br>Perception Since Baseline? | Any Changes in Vision or Light<br>Perception since Prior Physical<br>Examination |
|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Screening | Date9. (xx) | Yes/No | | |
| | | Baseline | Not Done : Reason | Yes/No | | |
| | | Day 1 | Date9. (xx) | Yes/No | Yes:Change/No | No |
| | | Day 7 | Date9. (xx) | Yes/No | _ | No |
| | | Day 28 | Date9. (xx) | Yes/No | | No |
| | | Month 3 | Date9. (xx) | Yes/No | | No |
| | | Month 6 | Date9. (xx) | Yes/No | | Yes: Changes |
| | | Month 12 or Early<br>Termination | Date9. (xx) | Yes/No | | Yes: Changes |

.....

Cohort 2 - 0.5 x 10<sup>6</sup> hRPC xxx--xxx

path\l\_program.sas date time

Protocol: JC-01

# Listing 16.2.8.9 Prior and Concomitant Medications

| | Subject | CM | Verbatim Term // | Start Date | Stop Date | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | ID | # | Preferred Drug Name | (Study Day) | (Study Day) | Dose | Units | Dose Form | Route | Frequency | Indication |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | 1 | Xxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Date9.(xx) | XXX | mg | Tablet | Oral | Daily | MH#, AE#,<br>injection<br>procedure |
| | | 2 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Ongoing | XXX | ug | Capsule | Oral | As Needed | • |
| | | 3 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Date9.(xx) | XX | ml | Suspension | Oral | Daily | |
| | | 4 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Ongoing | XXX | g | Ointment | Oral | Daily | |
| | | 5 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Ongoing | XX | Tablets | Tablet | Oral | Daily | |
| | | 6 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Date9.(xx) | XXX | Capsules | Capsule | Oral | Daily | |
| | | 7 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Ongoing | XXX | Puff | Aerosol | Oral | 2X a Day | |
| | | 8 | Xxxxxxxxxxxx // xxxxxxxxxxx | Date9.(xx) | Date9.(xx) | XXX | mg | Powder | Oral | Every Month | |

.....

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

path\l\_program.sas date time

Programmer Note: sort by CM # within each subject.

### Listing 16.2.8.10 Pregnancy Test

| Treatment Group | Subject<br>ID | Visit | Urine<br>Pregnancy<br>Collection Date<br>(Study Day) | Result | If Positive, Was a<br>Serum Test<br>Performed? | If Serum Test<br>Performed,<br>Result |
|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Screening<br>Baseline<br>Month 12 or Early<br>Termination | Date9. (xx) Date9. (xx) Date9. (xx) | Positive/Negative<br>Positive/Negative<br>Positive/Negative | Yes/No<br>Yes/No<br>Yes/No | Positive/Negative<br>Positive/Negative<br>Positive/Negative |

Not Done: Reason

path\l\_program.sas date time

Cohort 2 - 0.5 x 10<sup>6</sup> hRPC

Programmer Note: If NO marked for urine collection, include reason in "Urine Pregnancy Collection Date" column.

XXX--XXX

## Listing 16.2.8.11 PRA and DRA Antibody Test Results Received

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date (Study Day) | Sample Collected |
|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline Day 14 Day 28 Month 12 or Early Termination | Date9. (xx) Date9. (xx) Date9. (xx) Date9. (xx) | Yes/No<br>Yes/No<br>Yes/No |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | | | |

path\l\_program.sas date time

Programmer Note: If a panel/donor reactive antibody sample was not collected, please display "Not Done" and the reason in the "Collection Date/Time" column.

#### Listing 16.2.8.12 HLA Antibody Testing

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date (Study Day) | Result | Other HLA Antibody Testing<br>Results/Reason |
|---|---|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening<br>Baseline | Date9. (xx) | xxxxxx | |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening<br>Baseline | Date9. (xx)<br>Date9. (xx) | XXXXXX<br>XXXXXX | |

path\l\_program.sas date time

Programmer Note: If a HLA antibody testing sample was not collected, please display "Not Done" and the reason in the "Collection Date" column.

jCyte, Inc. Protocol: JC-01 Page 1 of x

# Listing 16.2.8.13 RP Gene Mutation Received

| Treatment Group | Subject<br>ID | Collection Date<br>(Study Day) | Sample Collected |
|---|---|---|---|
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX | Date9. (xx) Date9. (xx) Date9. (xx) | |
| | xxxxxx | | |

path\l\_program.sas date time

Programmer Note: For Other Row, show either Subject or Related under HLAA Typing Result column

## Listing 16.2.8.14.1 Slit Lamp Exam (OD) Part 1 of 2

| | Subject | | Exam Date (Study | у | Change from<br>Previous | 1 | Change from Previous | 1 | Change from Previous | | Change from Previous | l | Change from Previous |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | ID | Visit | Day) | Eyelids | Visit? | Eyelashes | Visit? | Conjunctiva | Visit? | Sclera | Visit? | Cornea | Visit? |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | Screening | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Baseline | Not Done:<br>Reason | Abnormal CS | Yes | Abnormal C | S Yes | Abnormal C | SYes | Abnormal C | S Yes | Abnormal C | S Yes |
| | | Day 1 | Date9.(xx) | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Day 2 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 3 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 7 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 14 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 21 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 28 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 2 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 3 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 4 | Date9.(xx) | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Month 5 | Date9.(xx) | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Month 6 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 9 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 12 or | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Early | . , | | | | | | | | | | |
| | | Termination | | | | | | | | | | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date

Programmer Note: If Slit Lamp Exam was not performed on left eye, please display "Not Done" and the reason in the "Exam Date" column.

Protocol No. JC-01

#### Listing 16.2.8.14.1 Slit Lamp Exam (OD) Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Exam<br>Date (Study<br>Day) | Anterior<br>Chamber<br>Flare | Change from<br>Previous<br>Visit? | ı<br>Iris | Change from<br>Previous<br>Visit? | Lens Status | Cataract<br>Type | Cataract<br>Grade | Clinically<br>Significant<br>Findings for<br>Grade? | Other Findings | Clinically<br>Significant<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | XXX | Screening | Date9.(xx) | 0 | | Normal | | Aphakic | Nuclear | +1 | Yes/No | Finding :<br>Abnoraml CS | Yes/No |
| | | Baseline | Not Done:<br>Reason | +1 | Yes | Abnormal C | SYes | Psedophakic | Cortical | +2 | Yes/No | | |
| | | Day 1 | Date9.(xx) | +1 | No | Abnormal<br>NCS | No | Phakic | Posterior | +3 | Yes/No | | |
| | | Day 2 | Date9.(xx) | +2 | | Normal | | Aphakic | Not<br>Applicable | +4<br>e | Yes/No | | |
| | | Day 3 | Date9.(xx) | +3 | | Normal | | Psedophakic | | +1 | Yes/No | | |
| | | Day 7 | Date9.(xx) | | | Normal | | Phakic | Cortical | +2 | Yes/No | | |
| | | Day 14 | Date9.(xx) | | | Normal | | Aphakic | Posterior | +3 | Yes/No | | |
| | | Day 21 | | | | Normal | | Psedophakic | | +4 | Yes/No | | |
| | | Day 28 | Date9.(xx) | +1 | | Normal | | Phakic | Cortical | +1 | Yes/No | | |
| | | Month 2 | Date9.(xx) | +4 | | Normal | | Aphakic | Posterior | +2 | Yes/No | | |
| | | Month 3 | Date9.(xx) | +1 | | Normal | | | Nuclear | +3 | Yes/No | | |
| | | Month 4 | Date9.(xx) | +3 | No | Abnormal<br>NCS | No | Phakic | Cortical | +4 | Yes/No | | |
| | | Month 5 | Date9.(xx) | +1 | No | Abnormal<br>NCS | No | Aphakic | Posterior | +1 | Yes/No | | |
| | | Month 6 | Date9.(xx) | +4 | | Normal | | Psedophakic | Nuclear | +2 | Yes/No | | |
| | | Month 9 | Date9.(xx) | | | Normal | | Phakic | Cortical | +3 | Yes/No | | |
| | | Month 12 or<br>Early<br>Termination | Date9.(xx) | | | Normal | | Aphakic | Posterior | +4 | Yes/No | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date

Programmer Note: If Slit Lamp Exam was not performed on left eye, please display "Not Done" and the reason in the "Exam Date" column. Programmer Note: Listing 16.2.8.14.2 will contain the same information for the other eye (OD).

### Listing 16.2.8.14.2 Slit Lamp Exam (OS) Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Exam Date (Study Day) | y<br>Eyelids | Change from<br>Previous<br>Visit? | Eyelashes | Change from<br>Previous<br>Visit? | n<br>Conjunctiva | Change from<br>Previous<br>Visit? | Sclera | Change from Previous Visit? | Cornea | Change from<br>Previous<br>Visit? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | xxxxxx | Screening | Date9.(xx) | • | | Normal | | Normal | | Normal | | Normal | |
| 10 <sup>6</sup> hRPC | | Baseline | Not Done:<br>Reason | Abnormal CS | Yes | Abnormal CS | S Yes | Abnormal C | SYes | Abnormal C | S Yes | Abnormal C | SYes |
| | | Day 1 | | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Day 2 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Day 3 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Day 7 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Day 14 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Day 21 | ( ) | | | Normal | | Normal | | Normal | | Normal | |
| • | | Day 28 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 2 | - ( ) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 3 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 4 | Date9.(xx) | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Month 5 | Date9.(xx) | Abnormal NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | Month 6 | Date9.(xx) | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 9 | Date9.(xx) | | | Normal | | Normal | | Normal | | Normal | |
| | | Month 12 or | \ / | | | Normal | | Normal | | Normal | | Normal | |
| | | Early<br>Termination | | | | | | | | | | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

Note: CS=Clinically Significant, NCS=Not Clinically Significant..

path\l\_program.sas date

Programmer Note: If Slit Lamp Exam was not performed on left eye, please display "Not Done" and the reason in the "Exam Date" column. Programmer Note: Listing 16.2.8.14.2 will contain the same information for the other eye (OS).

Protocol No. JC-01

## Listing 16.2.8.14.2 Slit Lamp Exam (OS) Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Exam<br>Date (Study<br>Day) | Anterior<br>Chamber<br>Flare | Change from<br>Previous<br>Visit? | ı<br>Iris | Change from<br>Previous<br>Visit? | Lens Status | Cataract<br>Type | Cataract<br>Grade | Clinically Significant Findings for Grade? | Other<br>Findings | Clinically<br>Significant<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - | | | • / | | | | | | | | | | |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | XXXXXX | Screening | Date9.(xx) | 0 | | Normal | | Aphakic | Nuclear | +1 | Yes/No | Finding:<br>Abnoraml CS | Yes/No |
| | | Baseline | Not Done:<br>Reason | +1 | Yes | Abnormal C | S Yes | Psedophakic | Cortical | +2 | Yes/No | | |
| | | Day 1 | Date9.(xx) | +1 | No | Abnormal<br>NCS | No | Phakic | Posterior | +3 | Yes/No | | |
| | | Day 2 | Date9.(xx) | +2 | | Normal | | Aphakic | Not<br>Applicable | +4 | Yes/No | | |
| | | Day 3 | Date9.(xx) | +3 | | Normal | | Psedophakic | | +1 | Yes/No | | |
| | | Day 7 | Date9.(xx) | | | Normal | | Phakic | Cortical | +2 | Yes/No | | |
| | | Day 14 | Date9.(xx) | +1 | | Normal | | Aphakic | Posterior | +3 | Yes/No | | |
| | | Day 21 | Date9.(xx) | | | Normal | | Psedophakic | Nuclear | +4 | Yes/No | | |
| | | Day 28 | Date9.(xx) | +1 | | Normal | | Phakic | Cortical | +1 | Yes/No | | |
| | | Month 2 | Date9.(xx) | +4 | | Normal | | Aphakic | Posterior | +2 | Yes/No | | |
| | | Month 3 | Date9.(xx) | +1 | | Normal | | Psedophakic | Nuclear | +3 | Yes/No | | |
| | | Month 4 | Date9.(xx) | +3 | No | Abnormal<br>NCS | No | Phakic | Cortical | +4 | Yes/No | | |
| | | Month 5 | Date9.(xx) | +1 | No | Abnormal<br>NCS | No | Aphakic | Posterior | +1 | Yes/No | | |
| | | Month 6 | Date9.(xx) | +4 | | Normal | | Psedophakic | Nuclear | +2 | Yes/No | | |
| | | Month 9 | Date9.(xx) | | | Normal | | Phakic | Cortical | +3 | Yes/No | | |
| | | Month 12 or<br>Early<br>Termination | Date9.(xx) | | | Normal | | Aphakic | Posterior | +4 | Yes/No | | |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date

Programmer Note: If Slit Lamp Exam was not performed on left eye, please display "Not Done" and the reason in the "Exam Date" column.
## Listing 16.2.8.15 Fundus Photography

| | | | | | OD | | OS |
|---|---|---|---|---|---|---|---|
| | | | Date | | If Right Eye Abnormal | _ | |
| | Subject | | Performed (Study | | Change from Previous | | If Left Eye Abnormal – |
| Treatment Group | ID | Visit | Day) | Results | Visit | Results | Change from Previous Visit |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | XXXXXX<br>XXX-XXX | Baseline<br>Baseline | Date9.(xx)<br>Not Done: Reason | Normal | | Normal | |
| | XXX-XXX | Baseline | Date9.(xx) | Abnormal CS:<br>Abnormality | Yes | Abnormal CS:Abnormality | Yes |
| | XXX-XXX | Baseline | Date9.(xx) | Abnormal NCS | Yes | Abnormal NCS | Yes |
| Cohort 2 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening | Date9.(xx) | | | | |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time

Programmer Note: If Fundus Photography was not performed, please display "Not Done" and the reason in the "Date Performed" column.

Listing 16.2.8.16 Intraocular Pressure (IOP)

| | C1.:4 | Measurement | | W T | IGN - Consider Desire | OD (B:-1-4) | OS (I -8) |
|---|---|---|---|---|---|---|---|
| _ | Subject | Date (Study | | Was a Tonopen | If No, Specify Device | OD (Right) | OS (Left) |
| Treatment Group | ID Visit | Day) | Time | Used? | Used | Mean IOP (mmHg) | Mean IOP (mmHg) |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx Baseline<br>Day 0 | Date9.(xx) Not done: Reason | Time5. | Yes/No | xxxxxxxx | xx | xx |
| | Day1 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 2 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 3 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 7 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 14 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 21 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Day 28 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 2 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 3 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 4 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 5 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 6 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 9 | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |
| | Month 12 or Early<br>Termination | Date9.(xx) | Time5. | Yes/No | xxxxxxxx | XX | XX |

Cohort 2 - 0.5 x 10<sup>6</sup> hRPC xxx--xxx Baseline Date9.(xx)

path\l\_program.sas date time

Programmer Note If an IOP measurement was not completed, please display "Not Done" and the reason in the "Measurement Date/Time" column.

### **Listing 16.2.8.17** B-Scan

| | | | | | Study | Eye | | Rig | ght Eye (OD) | | | | Left Eye (OS) | ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Measurem | | Injected Cells | | · | Abnormal, | | | | Abnormal, | | _ |
| | | | ent Date | | Visualized?if | • | | Change from | Pathology | Overall | | Change from | Pathology | Overall |
| Treatment | Subject | | (Study | | Yes, | Video | B-Scan | Previous | Result | Pathology | B-Scan | Previous | Result | Pathology |
| Group | ID | Visit | Day) | Time | Description | Taken? | Result | Visit? | Observed | Result | Result | Visit? | Observed | Result |
| Cohort 1 - 0.5<br>x 10 <sup>6</sup> hRPC | XXXXXX | Baseline | Date9.(xx) | Time5. | Yes:<br>Description/<br>No/NA | Yes/No/NA | Normal | Yes/No/NA | Retinal<br>Detachment | Good/Poor | Normal | Yes/No/NA | Retinal<br>Detachment | Good/Poor |
| | | Day 3 | Not done:<br>Reason | | | | | | | | | | | |
| | | Day 7 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Abnormal<br>CS:Abnormalit<br>y | Yes/No/NA | Irregular<br>Posterior<br>detachment | Good/Poor | CS:Abnorm Poster ality detachn | S:Abnorm Po<br>ality deta | Irregular<br>Posterior<br>detachment | Good/Poor |
| | | Month 3 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Abnormal<br>NCS | Yes/No/NA | | Good/Poor | Abnormal<br>NCS | Yes/No/NA | | Good/Poor |
| | | Month 6 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |
| | | Month 12 c<br>Early<br>Termination | or Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |
| Cohort 1 - 0.5<br>x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |
| x to inde | | Day 3 | Not done:<br>Reason | | | | | | | | | | | |
| | | Day 7 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Abnormal<br>CS:Abnormalit<br>y | Yes/No/NA | | Good/Poor | Abnormal<br>CS:Abnorm<br>ality | Yes/No/NA | | Good/Poor |
| | | Month 3 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Abnormal<br>NCS | Yes/No/NA | | Good/Poor | | Yes/No/NA | | Good/Poor |
| | | Month 6 | Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |
| | | Month 12 c<br>Early<br>Termination | or Date9.(xx) | Time5. | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date

Programmer Note: If B-Scan measurement was not completed, please display "Not Done" and the reason in the "Measurement Date/Time" column. Programmer Note Include description of abnormality and Clinically Significant information in "B-Scan Result" column.

# Listing 16.2.8.18 Dilated Funduscopic Examination Part 1 of 4

OD (Right)

| | | | | | - | | | <u> </u> | 2 (1118111) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Subject<br>ID | Visit | Time of<br>Dilator<br>Administrat<br>ion | Examination<br>Date (Study<br>Day) | Time of Examination | Vitreous<br>Exam Results | If Abnormal,<br>Change from<br>Previous Visit? | Vitreous Exam<br>Severity | Optic Nerve Exam | If Abnormal,<br>Change from<br>Previous Visit? | Optic Nerve Exam<br>Severity |
| Cohort 1 - 0.5 x 10 <sup>6</sup> hRPC | xxxxxx | Screening | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Baseline | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | ••••• | Day 1 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Severe | Abnormal CS:<br>Abnormality | Yes | Severe |
| | | Day 2 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Very Server | Abnormal NCS | No | Very Server |
| | | Day 3 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Day 7 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 14 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Day 21 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |
| | | Day 28 | Time5. | Date9. (xx) | Time5. | Not Done | | Mild | Not Done | | Mild |
| | | Month 2 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 3 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Mild | Abnormal CS:<br>Abnormality | Yes | Mild |
| | | Month 4 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Not Done | Abnormal NCS | No | Not Done |
| | | Month 5 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Month 6 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 9 | Time5. | Date9. (xx) | Time5. | Abnormal CS: | Yes | Mild | Abnormal CS: | Yes | Mild |
| | | | | ( ) | | Abnormality | | | Abnormality | | |
| | | Month 12 or<br>Early | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |

Cohort 2 - xxx--xxx 0.5 x 10<sup>6</sup> hRPC Termination

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant.

path\l program.sas date time

Protocol No. JC-01

#### **Listing 16.2.8.18 Dilated Funduscopic Examination** Part 2 of 4

| | | | | | OD (Right) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Time of | | | | If Abnormal, | | | | |
| | | | Dilator | Examination | Time of | | Change from | | | If Abnormal, Change | |
| Treatment | Subject | | | t Date (Study | Examination | Macula | Previous | Macula Exam | Peripheral Retina | from Previous Visit? | Peripheral Retina Exam |
| Group | ID | Visit | ion | Day) | | Exam Results | Visit? | Severity | Exam Results | | Severity |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | XXXXXX | Screening | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Baseline | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 1 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Severe | Abnormal CS: Abnormality | Yes | Severe |
| | | Day 2 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Very Server | Abnormal NCS | No | Very Server |
| | | Day 3 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Day 7 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 14 | Time5. | Date9. (xx) | Time5. | Abnormal CS: | Yes | Mild | Abnormal CS: | Yes | Mild |
| | | | | | | Abnormality | | | Abnormality | | |
| | | Day 21 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |
| | | Day 28 | Time5. | Date9. (xx) | Time5. | Not Done | | Mild | Not Done | | Mild |
| | | Month 2 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 3 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Month 4 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Not Done | Abnormal NCS | No | Not Done |
| | | Month 5 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Month 6 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 9 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Month 12 or<br>Early<br>Termination | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |

Cohort 2 - 0.5 x xxx--xxx

 $10^6 \, hRPC$ 

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant. path\l\_program.sas date

# Listing 16.2.8.18 Dilated Funduscopic Examination Part 3 of 4

OS(Left)

| Treatment<br>Group | Subject<br>ID | Visit | Time of Dilator<br>Administration | Examination<br>Date (Study<br>Day) | Time of<br>Examination | Vitreous<br>Exam Results | If Abnormal,<br>Change from<br>Previous Visit? | Vitreous Exam<br>Severity | Optic Nerve Exam | If Abnormal,<br>Change from<br>Previous Visit? | Optic Nerve Exam<br>Severity |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 - 0.5<br>x 10 <sup>6</sup> hRPC | xxxxxx | Screening | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Baseline | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 1 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Severe | Abnormal CS: Abnormality | Yes | Severe |
| | | Day 2<br>Day 3 | Time5.<br>Time5. | Date9. (xx)<br>Date9. (xx) | Time5.<br>Time5. | Abnormal NCS<br>Normal | No | Very Server<br>Mild | Abnormal NCS<br>Normal | No | Very Server<br>Mild |
| | | Day 7 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 14 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Day 21<br>Day 28 | Time5.<br>Time5. | Date9. (xx)<br>Date9. (xx) | Time5. | Abnormal NCS<br>Not Done | No | Moderate<br>Mild | Abnormal NCS<br>Not Done | No | Moderate<br>Mild |
| | | Month 2 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 3 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Month 4<br>Month 5 | Time5.<br>Time5. | Date9. (xx)<br>Date9. (xx) | Time5.<br>Time5. | Abnormal NCS<br>Normal | No | Not Done<br>Mild | Abnormal NCS<br>Normal | No | Not Done<br>Mild |
| | | Month 6 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 9 | Time5. | Date9. (xx) | Time5. | Abnormal CS: Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Month 12<br>or Early<br>Terminati<br>on | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |

Cohort 2 - 0.5 xxx--xxx x 10<sup>6</sup> hRPC

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant. path'l program.sas date time

Programmer Note: Sorting order is by Cohort #, subject ID, examination date (include unscheduled visits in the date sequence), and examination time.

# Protocol No. JC-01

### **Listing 16.2.8.18 Dilated Funduscopic Examination** Part 4 of 4

| | | | | | | | | | OS (Left) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Time of<br>Dilator | Examination | Time of<br>Examination | | If Abnormal,<br>Change from<br>Previous Visit? | | If Abnormal,<br>Change from | | |
| Treatment | Subject | | Administrat | Date (Study | | Macula | | Macula Exam | Peripheral Retina | Previous | Peripheral Retina |
| Group | ID | Visit | ion | Day) | | Exam Results | | Severity | Exam Results | Visit? | Exam Severity |
| Cohort 1 - 0.5 x<br>10 <sup>6</sup> hRPC | xxxxxx | Screening | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Baseline | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 1 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Severe | Abnormal CS:<br>Abnormality | Yes | Severe |
| | | Day 2 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Very Server | Abnormal NCS | No | Very Server |
| | | Day 3 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Day 7 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Day 14 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Day 21 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |
| | | Day 28 | Time5. | Date9. (xx) | Time5. | Not Done | | Mild | Not Done | | Mild |
| | | Month 2 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 3 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Mild | Abnormal CS: Abnormality | Yes | Mild |
| | | Month 4 | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Not Done | Abnormal NCS | No | Not Done |
| | | Month 5 | Time5. | Date9. (xx) | Time5. | Normal | | Mild | Normal | | Mild |
| | | Month 6 | Time5. | Date9. (xx) | Time5. | Not Done | | Moderate | Not Done | | Moderate |
| | | Month 9 | Time5. | Date9. (xx) | Time5. | Abnormal CS:<br>Abnormality | Yes | Mild | Abnormal CS:<br>Abnormality | Yes | Mild |
| | | Month 12 or<br>Early<br>Termination | Time5. | Date9. (xx) | Time5. | Abnormal NCS | No | Moderate | Abnormal NCS | No | Moderate |

Cohort 2 - 0.5 x xxx--xxx  $10^6 \, hRPC$ 

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant.

path\l program.sas date

Programmer Note: Sorting order is by Cohort #, subject ID, examination date (include unscheduled visits in the date sequence), and examination time.



Page 120/120